CLINICAL TRIAL: NCT03084796
Title: A 6-week, Multicenter, Randomized, Double-blind, Placebo and Active-controlled, Parallel Group, Dose-ranging Study to Evaluate the Efficacy and Safety of 4 Doses of CHF 5259 pMDI (HFA Glycopyrronium Bromide Via Pressurized Metered Dose Inhaler) in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A 6-week Dose Ranging Study of CHF 5259 pMDI in Subjects With Chronic Obstructive Pulmonary Disease
Acronym: GLIMMER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CCD-05993AA3-02
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: CHF 5259; Chronic Obstructive Pulmonary Disease (COPD); pMDI (pressurized metered dose inhaler); GLIMMER
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): CHF 5259 pMDI 6.25 μg, 1 inhalation twice daily (bid); (total daily dose [TDD] of CHF 5259 12.5 μg)
  Interventions: Drug: CHF 5259
- Treatment B (Experimental): CHF 5259 pMDI 12.5 μg, 1 inhalation bid; (TDD of CHF 5259: 25 μg)
  Interventions: Drug: CHF 5259
- Treatment C (Experimental): CHF 5259 pMDI 12.5 μg, 2 inhalations bid; (TDD of CHF 5259: 50 μg)
  Interventions: Drug: CHF 5259
- Treatment D (Experimental): CHF 5259 pMDI 25 μg, 2 inhalations bid; (TDD of CHF 5259: 100 μg)
  Interventions: Drug: CHF 5259
- Treatment E (Placebo Comparator): Placebo, 2 inhalations of CHF 5259 pMDI-matched Placebo bid;
  Interventions: Drug: Placebo
- Treatment F (Active Comparator): Tiotropium (TIO) 18 μg, SPIRIVA® HandiHaler®, 2 inhalations once daily (od) of the content of 1 capsule; (TDD of TIO: 18 μg)
  Interventions: Drug: Tiotropium Bromide 18 µg Inhalation Capsule

INTERVENTIONS:
Drug: CHF 5259 — Dose Response: Test one of four different doses of CHF 5259
  Arms: Treatment A; Treatment B; Treatment C; Treatment D
Drug: Placebo — Placebo Control
  Arms: Treatment E
Drug: Tiotropium Bromide 18 µg Inhalation Capsule — Active Control
  Other Names: SPIRIVA® HANDIHALER®
  Arms: Treatment F

SUMMARY:
The purpose of this study is to evaluate the dose-response of different doses of CHF 5259 pMDI on lung function and other clinical outcomes, to identify the optimal dose(s) in terms of benefit/ risk ratio for further development in the target subject population.

DETAILED DESCRIPTION:
This is a phase II, multicenter, randomized, double-blind, placebo and active controlled dose-ranging 6-arm parallel group study to identify the optimal dose of CHF 5259 pMDI (pressurized metered dose inhaler) with respect to lung function as well as other clinical efficacy and safety outcomes.

After a 2 week run-in period under rescue albuterol and background inhaled corticosteroid (ICS) as needed, patients were randomized to one of the 6 study treatment groups. Following randomization, subjects were assessed after 3 weeks and 6 weeks of study treatment at the study center. A follow-up phone was performed a week after the last visit.

During the study, daily symptoms, rescue and background medication use and compliance with the study drug were recorded in a subject diary. Treatment-Emergent Adverse Events (TEAEs) were assessed and recorded throughout the study. At screening and subsequent visits, subjects underwent physical and vital signs examinations, spirometry measurements, and 12-lead electrocardiogram (ECG). Symptoms and chronic obstructive pulmonary disease (COPD) health status were assessed through validated questionnaires. Routine hematology, blood chemistry, and pregnancy testing were performed before enrollment and at end of study. 24-hour (24-H) digital recording of ECGs (Holter) was performed before and after the first dose and just before the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 40 who have signed an Informed Consent Form prior to initiation of any study-related procedure.
* Subjects with a diagnosis of COPD (according to GOLD 2017 Global Strategy for the Diagnosis, Management and Prevention of COPD Report) at least 12 months before the screening visit.
* Current smokers or ex-smokers who quit smoking at least 6 months prior to screening visit, with a smoking history of at least 10 pack years
* A post-bronchodilator forced expiratory volume in the 1st second (FEV1) ≥50% and <80% of the predicted normal value and,
* a post-bronchodilator FEV1/ Forced Vital Capacity (FVC) < 0.7 at screening and
* a demonstrated reversibility to ipratropium defined as ΔFEV1 ≥ 5% over baseline 30-45 minutes after inhaling 4 puffs of ipratropium
* Subjects under regular COPD therapy for at least 2 months prior to screening with either inhaled long-acting muscarinic antagonist (LAMA), inhaled ICS/ long-acting β2-agonist (LABA), inhaled ICS + LAMA
* Symptomatic subjects at screening with a CAT score ≥10. This criterion must be confirmed at randomization
* Symptomatic subjects with a BDI focal score ≤ 10. This criterion must be confirmed at randomization
* A cooperative attitude and ability to demonstrate correct use of the inhalers and e-diary.

Exclusion Criteria:

* Pregnant or lactating women and all women physiologically capable of becoming pregnant UNLESS they are willing to use highly effective birth control methods
* Diagnosis of asthma or Asthma-COPD Overlap Syndrome (ACOS) as described in global initiative for asthma (GINA) Report 2016, history of allergic rhinitis or atopy (atopy which may raise contra-indications or impact the efficacy of the study treatment according to Investigator's judgment)
* COPD Exacerbations: a moderate or severe COPD exacerbation that has not resolved ≤14 days prior to screening and ≤30 days following the last dose of any oral/systemic corticosteroid or antibiotic (whichever comes last). A Moderate or Severe COPD exacerbation during the run-in period
* Use of antibiotics for a lower respiratory tract infection in the 4 weeks prior to screening or during run-in
* Subjects treated with non-cardio-selective β-blockers in the month preceding screening or during the run-in period
* Subjects treated with long-acting anti-histamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study, or if taken as needed
* Subjects requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia
* Known respiratory disorders other than COPD which may impact the efficacy of the study treatment according the Investigator's judgment.
* Subjects who have clinically significant cardiovascular condition
* Subjects who have a clinically significant abnormal 12-lead ECG that results in active medical problem which may impact the safety of the subject according to Investigator's judgement
* Subjects whose 12-lead ECG shows Fridericia corrected QT interval (QTcF) >450 ms for males or QTcF >470 ms for females at screening visit
* Medical diagnosis of narrow-angle glaucoma, clinically relevant prostatic hypertrophy or bladder neck obstruction that in the opinion of the Investigator would prevent use of anticholinergic agents
* History of hypersensitivity to M3 receptor antagonists, β2-adrenergic receptor agonist, corticosteroids or any of the excipients contained in any of the formulations used in the study which may raise contra-indications or impact the efficacy of the study treatment according to the Investigator's judgement
* Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease which may impact the efficacy or the safety of the study treatment according to Investigator's judgement
* Subjects with serum potassium levels <3.5 mEq/L (or 3.5 mmol/L) at screening
* Use of potent cytochrome P450 2D6 and 3A4 inhibitors within 4 weeks prior to screening
* Unstable or uncontrolled concurrent disease; fever, endocrine disease, gastrointestinal disease; neurological disease; hematological disease; autoimmune disorders, or other which may impact the feasibility of the results of the study according to Investigator's judgment
* History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening
* Subjects who have received an investigational drug within 1 month or 5 half-lives (whichever is greater) prior to screening visit, or have been previously randomized in this trial, or are currently participating in another clinical trial.
* Subjects who are mentally or legally incapacitated, or subjects accommodated in an establishment as a result of an official or judicial order.
* Subjects who have undergone major surgery in the 3 months prior to screening visit or have a planned surgery during the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kerwin, MD, Principal Investigator — Crisor LLC c/o Clinical Research Institute of Southern Oregon, Inc.
Locations (102):
- United States (102):
  - Chiesi Investigational Site, Birmingham, Alabama
  - Chiesi Investigational Site, Dothan, Alabama
  - Chiesi Investigational Site, Montgomery, Alabama
  - Chiesi Investigational Site, Flagstaff, Arizona
  - Chiesi Investigational Site, Glendale, Arizona
  - Chiesi Investigational Site, Phoenix, Arizona
  - Chiesi Investigational Site, Surprise, Arizona
  - Chiesi Investigational Site, Tempe, Arizona
  - Chiesi Investigational Site, Tucson, Arizona
  - Chiesi Investigational Site, Anaheim, California
  - Chiesi Investigational Site, Escondido, California
  - Chiesi Investigational Site, Fullerton, California
  - Clinical Trials Research, Lincoln, California
  - Chiesi Investigational Site, Long Beach, California
  - Chiesi Investigational Site, Los Angeles, California
  - Chiesi Investigational Site, Newport Beach, California
  - Chiesi Investigational Site, San Diego, California
  - Chiesi Investigational Site, Tustin, California
  - Chiesi Investigational Site, Westminster, California
  - Chiesi Investigational Site, Boulder, Colorado
  - Chiesi Investigational Site, Centennial, Colorado
  - Chiesi Investigational Site, Denver, Colorado
  - Chiesi Investigational Site, Lafayette, Colorado
  - Chiesi Investigational Site, Brandon, Florida
  - Chiesi Investigational Site, Clearwater, Florida
  - Chiesi Investigational Site, Daytona Beach, Florida
  - Chiesi Investigational Site, Edgewater, Florida
  - Chiesi Investigational Site, Hialeah, Florida
  - Chiesi Investigational Site, Kissimmee, Florida
  - Chiesi Investigational Site, Miami, Florida
  - Chiesi Investigational Site, Orlando, Florida
  - Chiesi Investigational Site, Panama City, Florida
  - Chiesi Investigational Site, Blue Ridge, Georgia
  - Chiesi Investigational Site, Dacula, Georgia
  - Chiesi Investigational Site, Duluth, Georgia
  - Chiesi Investigational Site, Lawrenceville, Georgia
  - Chiesi Investigational Site, Marietta, Georgia
  - Chiesi Investigational Site, Savannah, Georgia
  - Chiesi Investigational Site, Chicago, Illinois
  - Chiesi Investigational Site, Evansville, Indiana
  - Chiesi Investigational Site, Valparaiso, Indiana
  - Chiesi Investigational Site, Louisville, Kentucky
  - Chiesi Investigational Site, Crowley, Louisiana
  - Chiesi Investigational Site, Lake Charles, Louisiana
  - Chiesi Investigational Site, Lutherville, Maryland
  - Chiesi Investigational Site, Fall River, Massachusetts
  - Chiesi Investigational Site, Ann Arbor, Michigan
  - Chiesi Investigational Site, Farmington Hills, Michigan
  - Chiesi Investigational Site, Minneapolis, Minnesota
  - Chiesi Investigational Site, Saint Charles, Missouri
  - Chiesi Investigational Site, St Louis, Missouri
  - Chiesi Investigational Site, Missoula, Montana
  - Chiesi Investigational Site, Omaha, Nebraska
  - Chiesi Investigational Site, Las Vegas, Nevada
  - Chiesi Investigational Site, Summit, New Jersey
  - Chiesi Investigational Site, Albuquerque, New Mexico
  - Chiesi Investigational Site, The Bronx, New York
  - Chiesi Investigational Site, Charlotte, North Carolina
  - Chiesi Investigational Site, Gastonia, North Carolina
  - Chiesi Investigational Site, Hendersonville, North Carolina
  - Chiesi Investigational Site, Mooresville, North Carolina
  - Chiesi Investigational Site, Raleigh, North Carolina
  - Chiesi Investigational Site, Shelby, North Carolina
  - Chiesi Investigational Site, Wilmington, North Carolina
  - Chiesi Investigational Site, Winston-Salem, North Carolina
  - Chiesi Investigational Site, Cincinnati, Ohio
  - Chiesi Investigational Site, Columbus, Ohio
  - Clinical Research Solutions, Dayton, Ohio
  - Chiesi Investigational Site, Grove City, Ohio
  - Chiesi Investigational Site, Edmond, Oklahoma
  - Chiesi Investigational Site, Oklahoma City, Oklahoma
  - Chiesi Investigational Site, Medford, Oregon
  - Chiesi Investigational Site, Portland, Oregon
  - Chiesi Investigational Site, Philadelphia, Pennsylvania
  - Chiesi Investigational Site, East Providence, Rhode Island
  - Chiesi Investigational Site, Anderson, South Carolina
  - Chiesi Investigational Site, Charleston, South Carolina
  - Chiesi Investigational Site, Easley, South Carolina
  - Chiesi Investigational Site, Fort Mill, South Carolina
  - Chiesi Investigational Site, Gaffney, South Carolina
  - Chiesi Investigational Site, Greenville, South Carolina
  - Chiesi Investigational Site, Mt. Pleasant, South Carolina
  - Chiesi Investigational Site, Orangeburg, South Carolina
  - Chiesi Investigational Site, Rock Hill, South Carolina
  - Chiesi Investigational Site, Seneca, South Carolina
  - Chiesi Investigational Site, Spartanburg, South Carolina
  - Chiesi Investigational Site, Union, South Carolina
  - Chiesi Investigational Site, Rapid City, South Dakota
  - Chiesi Investigational Site, Franklin, Tennessee
  - Chiesi Investigational Site, Jackson, Tennessee
  - Chiesi Investigational Site, Knoxville, Tennessee
  - Chiesi Investigational Site, Tullahoma, Tennessee
  - Chiesi Investigational Site, Boerne, Texas
  - Chiesi Investigational Site, Cypress, Texas
  - Chiesi Investigational Site, New Braunfels, Texas
  - Chiesi Investigational Site, Sherman, Texas
  - Chiesi Investigational Site, Tomball, Texas
  - Chiesi Investigational Site, South Burlington, Vermont
  - Chiesi Investigational Site, Richmond, Virginia
  - Chiesi Investigational Site, Everett, Washington
  - Chiesi Investigational Site, Richland, Washington
  - Chiesi Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Tilert T, Dillon C, Paulose-Ram R, Hnizdo E, Doney B. Estimating the U.S. prevalence of chronic obstructive pulmonary disease using pre- and post-bronchodilator spirometry: the National Health and Nutrition Examination Survey (NHANES) 2007-2010. Respir Res. 2013 Oct 9;14(1):103. doi: 10.1186/1465-9921-14-103. PMID 24107140
- [Background] Mannino DM. COPD: epidemiology, prevalence, morbidity and mortality, and disease heterogeneity. Chest. 2002 May;121(5 Suppl):121S-126S. doi: 10.1378/chest.121.5_suppl.121s. PMID 12010839
- [Background] Tonnesen P. Smoking cessation and COPD. Eur Respir Rev. 2013 Mar 1;22(127):37-43. doi: 10.1183/09059180.00007212. PMID 23457163
- [Background] van Eerd EA, van der Meer RM, van Schayck OC, Kotz D. Smoking cessation for people with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2016 Aug 20;2016(8):CD010744. doi: 10.1002/14651858.CD010744.pub2. PMID 27545342
- [Background] Kew KM, Mavergames C, Walters JA. Long-acting beta2-agonists for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2013 Oct 15;2013(10):CD010177. doi: 10.1002/14651858.CD010177.pub2. PMID 24127118
- [Background] McGarvey L, Niewoehner D, Magder S, Sachs P, Tetzlaff K, Hamilton A, Korducki L, Bothner U, Vogelmeier C, Koch A, Ferguson GT. One-Year Safety of Olodaterol Once Daily via Respimat(R) in Patients with GOLD 2-4 Chronic Obstructive Pulmonary Disease: Results of a Pre-Specified Pooled Analysis. COPD. 2015;12(5):484-93. doi: 10.3109/15412555.2014.991864. Epub 2015 Feb 18. PMID 25692310
- [Background] Dahl R, Chung KF, Buhl R, Magnussen H, Nonikov V, Jack D, Bleasdale P, Owen R, Higgins M, Kramer B; INVOLVE (INdacaterol: Value in COPD: Longer Term Validation of Efficacy and Safety) Study Investigators. Efficacy of a new once-daily long-acting inhaled beta2-agonist indacaterol versus twice-daily formoterol in COPD. Thorax. 2010 Jun;65(6):473-9. doi: 10.1136/thx.2009.125435. PMID 20522841
- [Background] Keating GM. Tiotropium bromide inhalation powder: a review of its use in the management of chronic obstructive pulmonary disease. Drugs. 2012 Jan 22;72(2):273-300. doi: 10.2165/11208620-000000000-00000. PMID 22217233
- [Background] Casaburi R, Kukafka D, Cooper CB, Witek TJ Jr, Kesten S. Improvement in exercise tolerance with the combination of tiotropium and pulmonary rehabilitation in patients with COPD. Chest. 2005 Mar;127(3):809-17. doi: 10.1378/chest.127.3.809. PMID 15764761
- [Background] Kesten S, Casaburi R, Kukafka D, Cooper CB. Improvement in self-reported exercise participation with the combination of tiotropium and rehabilitative exercise training in COPD patients. Int J Chron Obstruct Pulmon Dis. 2008;3(1):127-36. doi: 10.2147/copd.s2389. PMID 18488436
- [Background] Karner C, Chong J, Poole P. Tiotropium versus placebo for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009285. doi: 10.1002/14651858.CD009285.pub2. PMID 22786525
- [Background] D'Urzo A, Ferguson GT, van Noord JA, Hirata K, Martin C, Horton R, Lu Y, Banerji D, Overend T. Efficacy and safety of once-daily NVA237 in patients with moderate-to-severe COPD: the GLOW1 trial. Respir Res. 2011 Dec 7;12(1):156. doi: 10.1186/1465-9921-12-156. PMID 22151296
- [Background] Kerwin E, Hebert J, Gallagher N, Martin C, Overend T, Alagappan VK, Lu Y, Banerji D. Efficacy and safety of NVA237 versus placebo and tiotropium in patients with COPD: the GLOW2 study. Eur Respir J. 2012 Nov;40(5):1106-14. doi: 10.1183/09031936.00040712. Epub 2012 Jul 26. PMID 23060624
- [Background] Beeh KM, Singh D, Di Scala L, Drollmann A. Once-daily NVA237 improves exercise tolerance from the first dose in patients with COPD: the GLOW3 trial. Int J Chron Obstruct Pulmon Dis. 2012;7:503-13. doi: 10.2147/COPD.S32451. Epub 2012 Jul 31. PMID 22973092
- [Background] Buhl R, Banerji D. Profile of glycopyrronium for once-daily treatment of moderate-to-severe COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:729-41. doi: 10.2147/COPD.S36001. Epub 2012 Oct 26. PMID 23118536
- [Background] Anthonisen NR, Connett JE, Enright PL, Manfreda J; Lung Health Study Research Group. Hospitalizations and mortality in the Lung Health Study. Am J Respir Crit Care Med. 2002 Aug 1;166(3):333-9. doi: 10.1164/rccm.2110093. PMID 12153966
- [Background] Michele TM, Pinheiro S, Iyasu S. The safety of tiotropium--the FDA's conclusions. N Engl J Med. 2010 Sep 16;363(12):1097-9. doi: 10.1056/NEJMp1008502. Epub 2010 Sep 8. No abstract available. PMID 20843240
- [Background] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213
- [Background] Wedzicha JA, Banerji D, Chapman KR, Vestbo J, Roche N, Ayers RT, Thach C, Fogel R, Patalano F, Vogelmeier CF; FLAME Investigators. Indacaterol-Glycopyrronium versus Salmeterol-Fluticasone for COPD. N Engl J Med. 2016 Jun 9;374(23):2222-34. doi: 10.1056/NEJMoa1516385. Epub 2016 May 15. PMID 27181606
- [Background] Yang IA, Fong KM, Sim EH, Black PN, Lasserson TJ. Inhaled corticosteroids for stable chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD002991. doi: 10.1002/14651858.CD002991.pub2. PMID 17443520
- [Background] Kew KM, Seniukovich A. Inhaled steroids and risk of pneumonia for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2014 Mar 10;2014(3):CD010115. doi: 10.1002/14651858.CD010115.pub2. PMID 24615270
- [Background] Yawn BP, Li Y, Tian H, Zhang J, Arcona S, Kahler KH. Inhaled corticosteroid use in patients with chronic obstructive pulmonary disease and the risk of pneumonia: a retrospective claims data analysis. Int J Chron Obstruct Pulmon Dis. 2013;8:295-304. doi: 10.2147/COPD.S42366. Epub 2013 Jun 27. PMID 23836970
- [Background] Rachelefsky GS, Liao Y, Faruqi R. Impact of inhaled corticosteroid-induced oropharyngeal adverse events: results from a meta-analysis. Ann Allergy Asthma Immunol. 2007 Mar;98(3):225-38. doi: 10.1016/S1081-1206(10)60711-9. PMID 17378253
- [Background] Roland NJ, Bhalla RK, Earis J. The local side effects of inhaled corticosteroids: current understanding and review of the literature. Chest. 2004 Jul;126(1):213-9. doi: 10.1378/chest.126.1.213. PMID 15249465
- [Background] Tashkin DP, Murray HE, Skeans M, Murray RP. Skin manifestations of inhaled corticosteroids in COPD patients: results from Lung Health Study II. Chest. 2004 Oct;126(4):1123-33. doi: 10.1016/S0012-3692(15)31287-3. PMID 15486373
- [Background] Crim C, Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Willits LR, Yates JC, Vestbo J. Pneumonia risk in COPD patients receiving inhaled corticosteroids alone or in combination: TORCH study results. Eur Respir J. 2009 Sep;34(3):641-7. doi: 10.1183/09031936.00193908. Epub 2009 May 14. PMID 19443528
- [Background] Crim C, Dransfield MT, Bourbeau J, Jones PW, Hanania NA, Mahler DA, Vestbo J, Wachtel A, Martinez FJ, Barnhart F, Lettis S, Calverley PM. Pneumonia risk with inhaled fluticasone furoate and vilanterol compared with vilanterol alone in patients with COPD. Ann Am Thorac Soc. 2015 Jan;12(1):27-34. doi: 10.1513/AnnalsATS.201409-413OC. PMID 25490706
- [Background] Pavord ID, Lettis S, Anzueto A, Barnes N. Blood eosinophil count and pneumonia risk in patients with chronic obstructive pulmonary disease: a patient-level meta-analysis. Lancet Respir Med. 2016 Sep;4(9):731-741. doi: 10.1016/S2213-2600(16)30148-5. Epub 2016 Jul 23. PMID 27460163
- [Background] Johnell O, Pauwels R, Lofdahl CG, Laitinen LA, Postma DS, Pride NB, Ohlsson SV. Bone mineral density in patients with chronic obstructive pulmonary disease treated with budesonide Turbuhaler. Eur Respir J. 2002 Jun;19(6):1058-63. doi: 10.1183/09031936.02.00276602. PMID 12108857
- [Background] Ferguson GT, Calverley PMA, Anderson JA, Jenkins CR, Jones PW, Willits LR, Yates JC, Vestbo J, Celli B. Prevalence and progression of osteoporosis in patients with COPD: results from the TOwards a Revolution in COPD Health study. Chest. 2009 Dec;136(6):1456-1465. doi: 10.1378/chest.08-3016. Epub 2009 Jul 6. PMID 19581353
- [Background] Loke YK, Cavallazzi R, Singh S. Risk of fractures with inhaled corticosteroids in COPD: systematic review and meta-analysis of randomised controlled trials and observational studies. Thorax. 2011 Aug;66(8):699-708. doi: 10.1136/thx.2011.160028. Epub 2011 May 20. PMID 21602540
- [Background] Suissa S, Kezouh A, Ernst P. Inhaled corticosteroids and the risks of diabetes onset and progression. Am J Med. 2010 Nov;123(11):1001-6. doi: 10.1016/j.amjmed.2010.06.019. Epub 2010 Oct 1. PMID 20870201
- [Background] Wang JJ, Rochtchina E, Tan AG, Cumming RG, Leeder SR, Mitchell P. Use of inhaled and oral corticosteroids and the long-term risk of cataract. Ophthalmology. 2009 Apr;116(4):652-7. doi: 10.1016/j.ophtha.2008.12.001. Epub 2009 Feb 25. PMID 19243828
- [Background] Miller DP, Watkins SE, Sampson T, Davis KJ. Long-term use of fluticasone propionate/salmeterol fixed-dose combination and incidence of cataracts and glaucoma among chronic obstructive pulmonary disease patients in the UK General Practice Research Database. Int J Chron Obstruct Pulmon Dis. 2011;6:467-76. doi: 10.2147/COPD.S14247. Epub 2011 Sep 16. PMID 22003292
- [Background] Andrejak C, Nielsen R, Thomsen VO, Duhaut P, Sorensen HT, Thomsen RW. Chronic respiratory disease, inhaled corticosteroids and risk of non-tuberculous mycobacteriosis. Thorax. 2013 Mar;68(3):256-62. doi: 10.1136/thoraxjnl-2012-201772. Epub 2012 Jul 10. PMID 22781123
- [Background] Aaron SD, Vandemheen KL, Fergusson D, Maltais F, Bourbeau J, Goldstein R, Balter M, O'Donnell D, McIvor A, Sharma S, Bishop G, Anthony J, Cowie R, Field S, Hirsch A, Hernandez P, Rivington R, Road J, Hoffstein V, Hodder R, Marciniuk D, McCormack D, Fox G, Cox G, Prins HB, Ford G, Bleskie D, Doucette S, Mayers I, Chapman K, Zamel N, FitzGerald M; Canadian Thoracic Society/Canadian Respiratory Clinical Research Consortium. Tiotropium in combination with placebo, salmeterol, or fluticasone-salmeterol for treatment of chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):545-55. doi: 10.7326/0003-4819-146-8-200704170-00152. Epub 2007 Feb 19. PMID 17310045
- [Background] Singh D, Brooks J, Hagan G, Cahn A, O'Connor BJ. Superiority of "triple" therapy with salmeterol/fluticasone propionate and tiotropium bromide versus individual components in moderate to severe COPD. Thorax. 2008 Jul;63(7):592-8. doi: 10.1136/thx.2007.087213. Epub 2008 Feb 1. PMID 18245142
- [Background] Hanania NA, Crater GD, Morris AN, Emmett AH, O'Dell DM, Niewoehner DE. Benefits of adding fluticasone propionate/salmeterol to tiotropium in moderate to severe COPD. Respir Med. 2012 Jan;106(1):91-101. doi: 10.1016/j.rmed.2011.09.002. Epub 2011 Oct 29. PMID 22040533
- [Background] Frith PA, Thompson PJ, Ratnavadivel R, Chang CL, Bremner P, Day P, Frenzel C, Kurstjens N; Glisten Study Group. Glycopyrronium once-daily significantly improves lung function and health status when combined with salmeterol/fluticasone in patients with COPD: the GLISTEN study, a randomised controlled trial. Thorax. 2015 Jun;70(6):519-27. doi: 10.1136/thoraxjnl-2014-206670. Epub 2015 Apr 3. PMID 25841237
- [Background] Siler TM, Kerwin E, Singletary K, Brooks J, Church A. Efficacy and Safety of Umeclidinium Added to Fluticasone Propionate/Salmeterol in Patients with COPD: Results of Two Randomized, Double-Blind Studies. COPD. 2016;13(1):1-10. doi: 10.3109/15412555.2015.1034256. Epub 2015 Oct 9. PMID 26451734
- [Background] Singh D, Papi A, Corradi M, Pavlisova I, Montagna I, Francisco C, Cohuet G, Vezzoli S, Scuri M, Vestbo J. Single inhaler triple therapy versus inhaled corticosteroid plus long-acting beta2-agonist therapy for chronic obstructive pulmonary disease (TRILOGY): a double-blind, parallel group, randomised controlled trial. Lancet. 2016 Sep 3;388(10048):963-73. doi: 10.1016/S0140-6736(16)31354-X. Epub 2016 Sep 1. PMID 27598678
- [Background] Chiesi Farmaceutici S.p.A. Randomised, double-blind, placebo-controlled, cross-over study to investigate the bronchodilator efficacy and safety after single and repeated administrations of different doses of glycopyrrolate via pMDI in moderate to severe COPD patients (GLYCO2). 2012 Jul 19; CCD-0916-CSR-0054.
- [Background] Novartis Pharmaceuticals Corporation. SEEBRI™ NEOHALER® US Prescribing Information. East Hanover, New Jersey; 2016 Jan.
- [Background] Boehringer Ingelheim Pharmaceuticals, Inc. SPIRIVA® HALER® US Prescribing Information. Ridgefield, Connecticut; 2016 Jan.
- [Background] Arievich H, Overend T, Renard D, Gibbs M, Alagappan V, Looby M, Banerji D. A novel model-based approach for dose determination of glycopyrronium bromide in COPD. BMC Pulm Med. 2012 Dec 8;12:74. doi: 10.1186/1471-2466-12-74. PMID 23217058
- [Background] LaForce C, Feldman G, Spangenthal S, Eckert JH, Henley M, Patalano F, D'Andrea P. Efficacy and safety of twice-daily glycopyrrolate in patients with stable, symptomatic COPD with moderate-to-severe airflow limitation: the GEM1 study. Int J Chron Obstruct Pulmon Dis. 2016 Jun 8;11:1233-43. doi: 10.2147/COPD.S100445. eCollection 2016. PMID 27354782
- [Background] Kerwin E, Siler TM, Korenblat P, White A, Eckert JH, Henley M, Patalano F, D'Andrea P. Efficacy and Safety of Twice-Daily Glycopyrrolate Versus Placebo in Patients With COPD: The GEM2 Study. Chronic Obstr Pulm Dis. 2016 Mar 28;3(2):549-559. doi: 10.15326/jcopdf.3.2.2015.0157. PMID 28848879
- [Background] Chiesi Farmaceutici S.p.A. A multinational, multicentre, randomised, double-blind, placebo-controlled, 2-way crossover study to evaluate the efficacy and safety of glycopyrrolate bromide administered via pMDI (CHF 5259), for the treatment of patients with chronic obstructive pulmonary disease. 2015 Nov 05; CCD-05993AA1-09.
- [Background] Mahler DA, Kerwin E, Ayers T, FowlerTaylor A, Maitra S, Thach C, Lloyd M, Patalano F, Banerji D. FLIGHT1 and FLIGHT2: Efficacy and Safety of QVA149 (Indacaterol/Glycopyrrolate) versus Its Monocomponents and Placebo in Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1068-79. doi: 10.1164/rccm.201505-1048OC. PMID 26177074
- [Background] Mahler DA, Gifford AH, Satti A, Jessop N, Eckert JH, D'Andrea P, Mota F, Banerjee R. Long-term safety of glycopyrrolate: A randomized study in patients with moderate-to-severe COPD (GEM3). Respir Med. 2016 Jun;115:39-45. doi: 10.1016/j.rmed.2016.03.015. Epub 2016 Mar 22. PMID 27215502
- [Background] Sharafkhaneh A, Majid H, Gross NJ. Safety and tolerability of inhalational anticholinergics in COPD. Drug Healthc Patient Saf. 2013;5:49-55. doi: 10.2147/DHPS.S7771. Epub 2013 Mar 8. PMID 23526112
- [Background] Chiesi Farmaceutici S.p.A. A multicentre, randomised, double-blind, active-controlled, 4-way cross-over study to evaluate the efficacy and safety of a free combination of 3 doses of glycopyrrolate with fixed combination beclomethasone dipropionate plus formoterol (FOSTER®) in a metered dose inhaler for the treatment of patients with chronic obstructive pulmonary disease (COPD). 2013 May 16; CCD-1106-PR-0066.
- [Background] Chiesi Farmaceutici S.p.A. Randomized, double-blind, active controlled, 3-arm parallel group, multi-national, multi-centre study to evaluate the cardiac safety of two doses of glycopyrrolate bromide (25µg and 50µg BID) delivered via HFA pMDI both combined with FOSTER® 100/6µg BID delivered via HFA pMDI versus FOSTER® 100/6µg BID delivered via HFA pMDI in patients with moderate to severe COPD. 2012 Jan 10; CCD-1107-PR-0067.
- [Background] Rennard S, Fogarty C, Reisner C, Fernandez C, Fischer T, Golden M, Rose ES, Darken P, Tardie G, Orevillo C. Randomized study of the safety, pharmacokinetics, and bronchodilatory efficacy of a proprietary glycopyrronium metered-dose inhaler in study patients with chronic obstructive pulmonary disease. BMC Pulm Med. 2014 Jul 16;14:118. doi: 10.1186/1471-2466-14-118. PMID 25027304
- [Background] Teva Respiratory LLC. QVAR® US Prescribing Information. Horsham, Pennsylvania; 2014 Jul.
- [Background] Mahler DA, Weinberg DH, Wells CK, Feinstein AR. The measurement of dyspnea. Contents, interobserver agreement, and physiologic correlates of two new clinical indexes. Chest. 1984 Jun;85(6):751-8. doi: 10.1378/chest.85.6.751. PMID 6723384
- [Background] Witek TJ Jr, Mahler DA. Minimal important difference of the transition dyspnoea index in a multinational clinical trial. Eur Respir J. 2003 Feb;21(2):267-72. doi: 10.1183/09031936.03.00068503a. PMID 12608440
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Jones PW, Tabberer M, Chen WH. Creating scenarios of the impact of COPD and their relationship to COPD Assessment Test (CAT) scores. BMC Pulm Med. 2011 Aug 11;11:42. doi: 10.1186/1471-2466-11-42. PMID 21835018
- [Background] Ellepola AN, Samaranayake LP. Inhalational and topical steroids, and oral candidosis: a mini review. Oral Dis. 2001 Jul;7(4):211-6. PMID 11575870
- [Background] Torres SR, Peixoto CB, Caldas DM, Silva EB, Akiti T, Nucci M, de Uzeda M. Relationship between salivary flow rates and Candida counts in subjects with xerostomia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Feb;93(2):149-54. doi: 10.1067/moe.2002.119738. PMID 11862202
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Hankinson JL, Kawut SM, Shahar E, Smith LJ, Stukovsky KH, Barr RG. Performance of American Thoracic Society-recommended spirometry reference values in a multiethnic sample of adults: the multi-ethnic study of atherosclerosis (MESA) lung study. Chest. 2010 Jan;137(1):138-45. doi: 10.1378/chest.09-0919. Epub 2009 Sep 9. PMID 19741060
- [Background] Hankinson JL, Bang KM. Acceptability and reproducibility criteria of the American Thoracic Society as observed in a sample of the general population. Am Rev Respir Dis. 1991 Mar;143(3):516-21. doi: 10.1164/ajrccm/143.3.516. PMID 2001060
- [Background] Boehringer Ingelheim Pharmaceuticals, Inc. ATROVENT® HFA US Prescribing Information. Ridgefield, Connecticut; 2012 Aug.
- [Background] Taylor J, Kotch A, Rice K, Ghafouri M, Kurland CL, Fagan NM, Witek TJ Jr; Ipratropium Bromide HFA Study Group. Ipratropium bromide hydrofluoroalkane inhalation aerosol is safe and effective in patients with COPD. Chest. 2001 Oct;120(4):1253-61. doi: 10.1378/chest.120.4.1253. PMID 11591569
- [Background] Singh D, Zhu CQ, Sharma S, Church A, Kalberg CJ. Daily variation in lung function in COPD patients with combined albuterol and ipratropium: results from a 4-week, randomized, crossover study. Pulm Pharmacol Ther. 2015 Apr;31:85-91. doi: 10.1016/j.pupt.2014.08.010. Epub 2014 Sep 6. PMID 25197005
- [Background] Beier J, van Noord J, Deans A, Brooks J, Maden C, Baggen S, Mehta R, Cahn A. Safety and efficacy of dual therapy with GSK233705 and salmeterol versus monotherapy with salmeterol, tiotropium, or placebo in a crossover pilot study in partially reversible COPD patients. Int J Chron Obstruct Pulmon Dis. 2012;7:153-64. doi: 10.2147/COPD.S26100. Epub 2012 Mar 5. PMID 22419863
- [Background] Leidy NK, Sexton CC, Jones PW, Notte SM, Monz BU, Nelsen L, Goldman M, Murray LT, Sethi S. Measuring respiratory symptoms in clinical trials of COPD: reliability and validity of a daily diary. Thorax. 2014 May;69(5):443-9. doi: 10.1136/thoraxjnl-2013-204428. Epub 2014 Mar 4. PMID 24595666
- [Background] Leidy NK, Murray LT, Monz BU, Nelsen L, Goldman M, Jones PW, Dansie EJ, Sethi S. Measuring respiratory symptoms of COPD: performance of the EXACT- Respiratory Symptoms Tool (E-RS) in three clinical trials. Respir Res. 2014 Oct 7;15(1):124. doi: 10.1186/s12931-014-0124-z. PMID 25287629
- [Background] Evidera. E-RS (EXACT-Respiratory Symptoms) User Manual (Version 3.0). Bethesda, Maryland; 2014 Oct.
- [Background] European Medicines Agency. Guideline on clinical investigation of medicinal products in the treatment of chronic obstructive pulmonary disease (COPD). c2012 Jun 21; EMA/CHMP/483572/2012.
- [Background] Donohue JF. Minimal clinically important differences in COPD lung function. COPD. 2005 Mar;2(1):111-24. doi: 10.1081/copd-200053377. PMID 17136971
- [Background] Mallinckrodt C, Roger J, Chuang-stein C, Molenberghs G, Lane PW, O'Kelly M, et al. Missing data: turning guidance into action. Stat Biopharm Res. 2013;5(4):369-82.
- [Background] Mallinckrodt CH, Kenward MG. Conceptual Considerations regarding Endpoints, Hypotheses, and Analyses for Incomplete Longitudinal Clinical Trial Data. Drug Inf J. 2009; 43(4): 449-58.
- [Background] National Research Council (US) Panel on Handling Missing Data in Clinical Trials. The Prevention and Treatment of Missing Data in Clinical Trials. Washington (DC): National Academies Press (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK209904/ PMID 24983040
- [Background] Leuchs AK, Zinserling J, Brandt A, Wirtz D, Benda N. Choosing Appropriate Estimands in Clinical Trials. Ther Innov Regul Sci. 2015 Jul;49(4):584-592. doi: 10.1177/2168479014567317. PMID 30222440
- [Background] Edwards D, Berry JJ. The efficiency of simulation-based multiple comparisons. Biometrics. 1987 Dec;43(4):913-28. PMID 3427176
- [Result] Kerwin E, Feldman G, Pearle J, De La Cruz L, Edwards M, Beaudot C, Georges G. Efficacy and Safety of Inhaled Glycopyrronium Bromide in COPD: A Randomized, Parallel Group, Dose-Ranging Study (GLIMMER). COPD. 2021 Apr;18(2):181-190. doi: 10.1080/15412555.2021.1894111. Epub 2021 Mar 12. PMID 33709856
- See also: From the Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2017. — https://goldcopd.org/wp-content/uploads/2017/02/wms-GOLD-2017-FINAL.pdf
- See also: Chiesi Respiratory — https://www.chiesi.com/en/air/
- See also: Chiesi Farmaceutici is the first company to submit a marketing authorisation application to the European Medicine Agency for a Triple Combination for the treatment of COPD — https://www.chiesi.com/en/chiesi-farmaceutici-is-the-first-company-to-submit-a-marketing-authorisation-application-to-the-european-medicine-agency-for-a-triple-combination-for-the-treatment-of-copd-
- See also: Glycopyrronium bromide — https://en.wikipedia.org/wiki/Glycopyrronium_bromide
- See also: American Thoracic Society: Baseline Dyspnea Index (BDI) & Transition Dyspnea Index (TDI). — http://www.thoracic.org/members/assemblies/assemblies/srn/questionaires/bdi-tdi.php
- See also: American Thoracic Society: COPD Assessment Test (CAT). — http://www.thoracic.org/members/assemblies/assemblies/srn/questionaires/copd.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: CHF 5259 pMDI Dose 1, 12.5 μg TDD
  CHF 5259 Dose Response: Test one of four different doses of CHF 5259
- Treatment B: CHF 5259 pMDI Dose 2, 25 μg TDD
  CHF 5259 Dose Response: Test one of four different doses of CHF 5259
- Treatment C: CHF 5259 pMDI Dose 3, 50 μg TDD
  CHF 5259 Dose Response: Test one of four different doses of CHF 5259
- Treatment D: CHF 5259 pMDI Dose 4, 100 μg TDD
  CHF 5259 Dose Response: Test one of four different doses of CHF 5259
- Treatment E: Placebo Control
  Placebo: Placebo Control
- Treatment F: Tiotropium Bromide inhalation powder, 18 µg TDD
  Tiotropium Bromide Active Control, 18 µg Inhalation Capsule
Period: Overall Study
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Started | 121 | 123 | 122 | 123 | 121 | 123
Completed | 114 | 113 | 110 | 119 | 110 | 116
Not Completed | 7 | 10 | 12 | 4 | 11 | 7
Not completed — Adverse Event | 4 | 5 | 6 | 2 | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5 | 2 | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 3 | 1
Not completed — Randomization error | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients male or female, aged ≥ 40 years with a diagnosis of COPD at least 12 months before the screening visit, who were current smokers or ex-smokers who had quit smoking at least 6 months prior to the screening visit, with a smoking history of at least 10 pack-years. Study inclusion and exclusion criteria are presented in the study protocol section.
Groups:
- Treatment A: CHF 5259 pMDI, 6.25 μg, 1 inhalation bid; 12.5 μg TDD
  CHF 5259 Dose Response: Test one of 4 different doses of CHF 5259
- Treatment B: CHF 5259 pMDI 12.5 μg, 1 inhalation bid; 25 μg TDD
  CHF 5259 Dose Response: Test one of 4 different doses of CHF 5259
- Treatment C: CHF 5259 pMDI 12.5 μg, 2 inhalations bid; 50 μg TDD
  CHF 5259 Dose Response: Test one of 4 different doses of CHF 5259
- Treatment D: CHF 5259 pMDI 25 μg, 2 inhalations bid; 100 μg TDD
  CHF 5259 Dose Response: Test one of 4 different doses of CHF 5259
- Treatment E: Placebo 2 inhalations of CHF 5259 pMDI-matched Placebo bid
  Placebo: Placebo Control
- Treatment F: Tiotropium Bromide inhalation powder, 18 μg, SPIRIVA® HandiHaler®, 2 inhalations od of the content of 1 capsule; 18 µg TDD
  Tiotropium Bromide Active Control, 18 µg Inhalation Capsule
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F | Total
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123 | 732
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.13) | 65.3 (9.10) | 65.3 (8.16) | 64.9 (9.11) | 64.9 (9.25) | 63.8 (9.55) | 64.7 (9.05)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 59 | 53 | 56 | 62 | 60 | 62 | 352
  65-84 years | 60 | 68 | 65 | 60 | 58 | 59 | 370
  > 85 years | 2 | 2 | 0 | 1 | 3 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 68 | 67 | 65 | 52 | 57 | 367
  Male | 63 | 55 | 54 | 58 | 69 | 66 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 12 | 11 | 5 | 7 | 51
  Not Hispanic or Latino | 114 | 114 | 109 | 112 | 115 | 116 | 680
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 10 | 14 | 12 | 10 | 69
  White | 107 | 110 | 107 | 108 | 104 | 110 | 646
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 4 | 1 | 1 | 2 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 123 | 121 | 123 | 121 | 123 | 732
Weight [Mean (Standard Deviation); unit: kg] | 81.81 (20.64) | 83.82 (19.33) | 82.12 (22.70) | 84.23 (22.41) | 84.43 (21.82) | 80.67 (17.40) | 82.85 (20.77)
Height [Mean (Standard Deviation); unit: cm] | 168.95 (8.76) | 169.38 (9.74) | 169.21 (9.67) | 168.17 (9.57) | 169.34 (9.56) | 169.53 (9.67) | 169.10 (9.48)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.67 (7.05) | 29.13 (5.98) | 28.52 (6.77) | 29.62 (6.73) | 29.26 (6.49) | 28.05 (5.54) | 28.88 (6.45)
Time since first diagnosis of COPD [Median (Full Range); unit: months] | 92.80 [14.9 to 337.2] | 99.60 [18.0 to 332.8] | 97.40 [13.6 to 370.5] | 94.00 [12.9 to 349.6] | 103.40 [18.2 to 380.4] | 74.40 [12.2 to 335.8] | 94.55 [12.2 to 380.4]
Age at first diagnosis of COPD [Mean (Standard Deviation); unit: years] | 54.98 (9.31) | 55.45 (9.29) | 55.38 (8.46) | 56.40 (9.41) | 55.12 (8.85) | 55.65 (10.19) | 55.50 (9.25)
COPD medication category at study entry [Count of Participants; unit: Participants]
  Inhaled LAMA | 24 | 22 | 31 | 22 | 25 | 27 | 151
  Inhaled ICS and LABA (free combination) | 3 | 0 | 0 | 1 | 0 | 2 | 6
  Inhaled ICS/LABA (fixed combination) | 77 | 89 | 74 | 92 | 78 | 81 | 491
  Inhaled ICS and LAMA | 0 | 1 | 2 | 1 | 2 | 2 | 8
  Inhaled ICS+LABA+LAMA (free or fixed combination) | 11 | 3 | 11 | 6 | 13 | 8 | 52
  Inhaled LABA/LAMA (fixed combination) | 6 | 8 | 3 | 1 | 3 | 3 | 24
Smoking habits [Count of Participants; unit: Participants]
  Current smoker | 61 | 59 | 59 | 68 | 55 | 67 | 369
  Ex-smoker | 60 | 64 | 62 | 55 | 66 | 56 | 363
Duration of smoking [Mean (Standard Deviation); unit: years] | 42.19 (9.74) | 42.98 (9.86) | 40.71 (10.46) | 42.78 (10.44) | 41.34 (10.39) | 40.79 (10.83) | 41.80 (10.30)
Number of pack-years [Median (Full Range); unit: pack-years] — A pack-year is a term used to describe the approximate number of cigarettes a person has smoked over time. 1 One pack-year equals 20 manufactured cigarettes smoked per day for one year.
  pack-years | 45.0 [11 to 132] | 49.0 [10 to 135] | 45.0 [10 to 159] | 45.0 [11 to 128] | 45.0 [10 to 150] | 43.0 [10 to 128] | 45.0 [10 to 159]
FEV1 (L) at baseline [Mean (Standard Deviation); unit: litres] — Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath during the first second (FEV1).
  litres | 1.440 (0.432) | 1.428 (0.439) | 1.434 (0.472) | 1.420 (0.419) | 1.415 (0.433) | 1.443 (0.487) | 1.430 (0.446)
FVC at baseline [Mean (Standard Deviation); unit: litres] — Forced vital capacity (FVC) is the maximal volume of gas that can be exhaled from full inhalation by exhaling as forcefully and rapidly as possible.
  litres | 2.717 (0.754) | 2.719 (0.775) | 2.669 (0.725) | 2.630 (0.719) | 2.683 (0.736) | 2.746 (0.809) | 2.694 (0.752)
IC at baseline [Mean (Standard Deviation); unit: litres] — Inspiratory capacity (IC) is the amount of air taken in during a deep breath, without hesitation, after a normal, relaxed expiration. IC is decreased in obstructive lung diseases.
  litres | 2.020 (0.622) | 2.065 (0.533) | 2.089 (0.683) | 2.066 (0.572) | 2.053 (0.628) | 2.175 (0.624) | 2.078 (0.612)
BDI focal scores at randomization [Mean (Standard Deviation); unit: scores on a scale] — Baseline Dyspnea Index (BDI): a validated, interviewer-administered rating of severity of dyspnea. It provides a multidimensional measurement of dyspnea evoked in activities of daily living, in symptomatic individuals during the last 2 weeks. BDI consists of 24 items (3 domains: Functional Impairment, Magnitude of Task, and Magnitude of Effort), each rated on a 5-point scale from 0 (very severe impairment) to 4 (no impairment), with a total score ranging from 0-12. Only patients with a BDI focal score ≤10 at screening, and at randomization were eligible for enrolment into the current trial.
  scores on a scale | 5.6 (1.88) | 5.9 (1.87) | 5.8 (1.77) | 5.8 (1.63) | 6.1 (1.43) | 5.7 (1.59) | 5.8 (1.71)
CAT total score at randomization [Mean (Standard Deviation); unit: scores on a scale] — COPD Assessment Test (CAT) is a patient-completed validated questionnaire. It measures the global impact of COPD on a patient's life in an objective way and monitors changes over time. CAT consists of eight items scored on a scale of 1 to 5, with a total score range of 0-40; a higher score denotes a more severe impact of COPD on a patient's life. Only patients with a CAT score ≥10 at screening and at randomisation were eligible for enrolment into the current trial.
  scores on a scale | 19.6 (5.60) | 19.2 (5.65) | 19.2 (5.83) | 20.0 (5.49) | 19.3 (5.73) | 20.3 (6.48) | 19.6 (5.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FEV1 AUC(0-12h) Normalized by Time at Week 6
Description: Change from baseline in FEV1 AUC(0-12h), normalized by time, at the end of treatment (Week 6).
  Spirometry, used to measure FEV1, was performed according to internationally accepted standards. The AUC for FEV1 at Week 6 of treatment was calculated by using the linear trapezoidal rule, based on the changes in FEV1 from the baseline values, and divided by the observation time (12 hours).
  Definitions:
  AUC=Area under the curve; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); FEV1=Forced expiratory volume in the 1st second; FEV1 AUC(0-12h)=Mean FEV1 after inhalation, measured at prespecified times for up to 12-h observation period (0-12 h), normalized by time;
Time Frame: Baseline, Week 6
Population: Intention to treat:
  All randomized patients who received at least one dose of the study treatment and with at least one available evaluation of efficacy after baseline (primary or secondary efficacy variables).
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 113 | 111 | 108 | 118 | 109 | 114
Litres | 0.070 [0.034 to 0.106] | 0.118 [0.082 to 0.155] | 0.153 [0.116 to 0.190] | 0.147 [0.111 to 0.183] | 0.002 [-0.035 to 0.039] | 0.213 [0.177 to 0.250]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison groups were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates. Adjusted for multiplicity based on the parametric simulation method by Edwards and Berry; Test type: Superiority; p = 0.037, Mixed Models Analysis; Mean Difference (Final Values) = 0.068, 95% CI 2-sided [0.003 to 0.132]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Comparison treatment groups were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis for was performed as described for the statistical analysis 1 for this outcome measure. Adjusted for multiplicity based on the parametric simulation method by Edwards and Berry; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.116, 95% CI 2-sided [0.051 to 0.181]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Comparison treatment groups were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis for was performed as described for the statistical analysis 1 for this outcome measure. Adjusted for multiplicity based on the parametric simulation method by Edwards and Berry; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.151, 95% CI 2-sided [0.086 to 0.216]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Comparison treatment groups were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis for was performed as described for the statistical analysis 1 for this outcome measure. Adjusted for multiplicity based on the parametric simulation method by Edwards and Berry; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.145, 95% CI 2-sided [0.081 to 0.209]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison treatment groups were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.211, 95% CI 2-sided [0.159 to 0.263]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison treatment groups were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.003 to 0.100]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Comparison treatment groups were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.083, 95% CI 2-sided [0.031 to 0.135]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Comparison treatment groups were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [0.026 to 0.128]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Comparison treatment groups were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD. Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p = 0.189, Mixed Models Analysis; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.017 to 0.087]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Comparison treatment groups were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p = 0.273, Mixed Models Analysis; Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.023 to 0.080]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Comparison treatment groups were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Analyzed using a linear mixed model for repeated measures (MMRM) including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West)" and smoking status at screening as fixed effects, and the baseline value and baseline by visit interaction as covariates; Test type: Superiority; p = 0.813, Mixed Models Analysis; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.058 to 0.045]

2. Secondary Outcome: Change From Baseline in FEV1 AUC(0-12h) Normalized by Time on Day 1
Description: Change from baseline in FEV1 AUC(0-12h), normalized by time, on Day 1.
  Spirometry, used to measure FEV1, was performed according to internationally accepted standards. The AUC for FEV1 on Day 1 of treatment was calculated by using the linear trapezoidal rule, based on the changes in FEV1 from the baseline values, and divided by the observation time (12 hours).
  Definitions:
  AUC=Area under the curve; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); Day 1=Day of the first dose of randomized study drug at Visit 2 (Week 0); FEV1=Forced expiratory volume in the 1st second; FEV1 AUC(0-12h)=Mean FEV1 after inhalation, measured at prespecified times for up to 12-h observation period (0-12 h), normalized by time;
Time Frame: Baseline, Day 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 120 | 121 | 121 | 122
Litres | 0.067 [0.041 to 0.093] | 0.086 [0.060 to 0.111] | 0.135 [0.109 to 0.161] | 0.149 [0.123 to 0.175] | 0.009 [-0.017 to 0.035] | 0.192 [0.166 to 0.218]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model for repeated measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [0.022 to 0.095]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [0.040 to 0.113]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.126, 95% CI 2-sided [0.089 to 0.163]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [0.104 to 0.177]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.183, 95% CI 2-sided [0.147 to 0.220]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p = 0.322, Mixed Models Analysis; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.018 to 0.055]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.067, 95% CI 2-sided [0.031 to 0.104]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.045 to 0.118]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD. Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [0.013 to 0.086]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [0.027 to 0.100]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 for this outcome measure; Test type: Superiority; p = 0.443, Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.022 to 0.051]

3. Secondary Outcome: Change From Baseline in FEV1 AUC(0-4h) Normalized by Time on Day 1 and at Week 6
Description: Change from baseline in FEV1 AUC(0-4h), normalized by time on Day 1 of treatment (Week 0).
  Spirometry, used to measure FEV1, was performed according to internationally accepted standards. The AUC for FEV1 on Day 1 and at Week 6 of treatment was calculated by using the linear trapezoidal rule, based on the changes in FEV1 from the baseline values, and divided by the observation time (4 hours).
  Definitions:
  AUC=Area under the curve; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); Day 1=Day of the first dose of randomized study drug at Visit 2 (Week 0); FEV1=Forced expiratory volume in the 1st second; FEV1 AUC(0-4h)=Mean FEV1 after inhalation, measured at prespecified times for up to 4-h observation period (0-4h), normalized by time;
Time Frame: Baseline, Day 1, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Day 1 | 0.101 [0.077 to 0.125] | 0.115 [0.091 to 0.139] | 0.173 [0.149 to 0.196] | 0.190 [0.166 to 0.214] | 0.030 [0.006 to 0.053] | 0.194 [0.170 to 0.218]
  Week 6: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  Week 6 | 0.116 [0.078 to 0.154] | 0.157 [0.118 to 0.195] | 0.198 [0.159 to 0.237] | 0.204 [0.167 to 0.242] | 0.024 [-0.015 to 0.062] | 0.253 [0.215 to 0.291]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Day 1 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model for repeated measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.072, 95% CI 2-sided [0.038 to 0.105]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Day 1 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.086, 95% CI 2-sided [0.052 to 0.119]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Day 1 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.143, 95% CI 2-sided [0.109 to 0.177]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Day 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.160, 95% CI 2-sided [0.127 to 0.194]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Day 1 Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.164, 95% CI 2-sided [0.131 to 0.198]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Day 1 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.418, Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.020 to 0.048]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Day 1 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [0.038 to 0.105]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Day 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [0.055 to 0.122]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Day 1 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [0.024 to 0.091]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Day 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [0.041 to 0.108]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Day 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.308, Mixed Models Analysis; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.016 to 0.051]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.092, 95% CI 2-sided [0.038 to 0.147]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Analyzed, using linear mixed model repeated measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.133, 95% CI 2-sided [0.079 to 0.188]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [0.120 to 0.229]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.181, 95% CI 2-sided [0.127 to 0.235]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; Week 6 Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.229, 95% CI 2-sided [0.175 to 0.284]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; Week 6 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.141, Mixed Models Analysis; Mean Difference (Final Values) = 0.041, 95% CI 2-sided [-0.013 to 0.095]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; Week 6 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.028 to 0.137]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; Week 6 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [0.035 to 0.142]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; Week 6 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.137, Mixed Models Analysis; Mean Difference (Final Values) = 0.041, 95% CI 2-sided [-0.013 to 0.096]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; Week 6 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.082, Mixed Models Analysis; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.006 to 0.101]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; Week 6 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.823, Mixed Models Analysis; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.048 to 0.060]

4. Secondary Outcome: Change From Baseline in FEV1 Peak(0-4h) at Day 1 and Week 6
Description: Change from baseline in FEV1 peak(0-4h) (L) on Day 1 and at Week 6.
  Peak FEV1 is defined as the maximum FEV1 observed in the first 4 hours after dose of study medication.
  Definitions:
  Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); Day 1=Day of the first dose of randomized study drug at Visit 2 (Week 0); FEV1=Forced expiratory volume in the 1st second; Peak(0-4h)=Maximum FEV1 between 0 and 4 h.
Time Frame: Baseline, Day 1, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Day 1 | 0.197 [0.170 to 0.224] | 0.211 [0.183 to 0.238] | 0.260 [0.233 to 0.287] | 0.288 [0.261 to 0.315] | 0.136 [0.109 to 0.163] | 0.299 [0.272 to 0.326]
  Week 6: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  Week 6 | 0.212 [0.171 to 0.253] | 0.255 [0.214 to 0.296] | 0.305 [0.263 to 0.346] | 0.301 [0.260 to 0.341] | 0.143 [0.102 to 0.185] | 0.356 [0.315 to 0.397]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Day 1 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [0.022 to 0.100]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [0.036 to 0.113]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.085 to 0.163]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.152, 95% CI 2-sided [0.113 to 0.190]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.001, MMRM; Mean Difference (Final Values) = 0.163, 95% CI 2-sided [0.124 to 0.202]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 0.485, Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.025 to 0.052]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [0.025 to 0.102]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [0.053 to 0.130]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [0.011 to 0.088]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.077, 95% CI 2-sided [0.039 to 0.116]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; p = 0.157, Mixed Models Analysis; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.011 to 0.066]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.021, Mixed Models Analysis; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [0.011 to 0.128]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.053 to 0.170]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.162, 95% CI 2-sided [0.103 to 0.220]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.157, 95% CI 2-sided [0.099 to 0.215]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.213, 95% CI 2-sided [0.154 to 0.271]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.149, Mixed Models Analysis; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.015 to 0.101]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.092, 95% CI 2-sided [0.034 to 0.151]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [0.031 to 0.146]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.096, Mixed Models Analysis; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [-0.009 to 0.108]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.122, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [-0.012 to 0.103]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.886, Mixed Models Analysis; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.062 to 0.054]

5. Secondary Outcome: Change From Baseline in FVC AUC(0-12h), Normalized by Time on Day 1 and at Week 6
Description: Change from baseline in FVC AUC(0-12h), normalized by time, on Day 1 and at the end of treatment (Week 6).
  Spirometry, used to measure FVC, was performed according to internationally accepted standards. The AUC for FVC was calculated by using the linear trapezoidal rule, based on the changes in FVC from the baseline values, and divided by the observation time (4 hours).
  Definitions:
  AUC=Area under the curve; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); Day 1=Day of the first dose of randomized study drug at Visit 2 (Week 0); FVC=Forced Vital Capacity; FVC AUC(0-12h)=Mean FVC after inhalation, measured at prespecified times for up to 12-h observation period (0-12 h), normalized by time;
Time Frame: Baseline, Day 1, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Day 1: number analyzed (Participants) | 121 | 123 | 120 | 121 | 121 | 122
  Day 1 | 0.086 [0.039 to 0.133] | 0.133 [0.086 to 0.180] | 0.195 [0.148 to 0.242] | 0.220 [0.173 to 0.267] | 0.011 [-0.036 to 0.058] | 0.305 [0.258 to 0.351]
  Week 6: number analyzed (Participants) | 113 | 111 | 108 | 118 | 109 | 114
  Week 6 | 0.084 [0.026 to 0.142] | 0.145 [0.087 to 0.203] | 0.190 [0.131 to 0.249] | 0.184 [0.127 to 0.241] | -0.029 [-0.087 to 0.030] | 0.298 [0.240 to 0.355]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = 0.074, 95% CI 2-sided [0.008 to 0.141]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [0.055 to 0.188]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.184, 95% CI 2-sided [0.117 to 0.250]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.208, 95% CI 2-sided [0.142 to 0.275]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.293, 95% CI 2-sided [0.227 to 0.360]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 0.161, Mixed Models Analysis; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [-0.019 to 0.113]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.109, 95% CI 2-sided [0.043 to 0.176]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.134, 95% CI 2-sided [0.068 to 0.201]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = 0.062, 95% CI 2-sided [-0.004 to 0.128]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.021 to 0.153]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; p = 0.465, Mixed Models Analysis; Mean Difference (Final Values) = 0.025, 95% CI 2-sided [-0.042 to 0.091]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 12]; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.030 to 0.195]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.173, 95% CI 2-sided [0.091 to 0.256]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.219, 95% CI 2-sided [0.136 to 0.302]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.213, 95% CI 2-sided [0.131 to 0.295]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p < 0.001, McNemar; Mean Difference (Final Values) = 0.326, 95% CI 2-sided [0.244 to 0.409]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.144, Mixed Models Analysis; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [-0.021 to 0.143]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = 0.107, 95% CI 2-sided [0.024 to 0.189]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.019 to 0.182]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.280, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [-0.037 to 0.128]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.342, Mixed Models Analysis; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.042 to 0.121]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.886, Mixed Models Analysis; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.088 to 0.076]

6. Secondary Outcome: Change From Baseline in FVC AUC(0-4h) Normalized by Time on Day 1 and at Week 6
Description: Change from baseline in FVC AUC(0-4h), normalized by time, on Day 1 and at the end of treatment (Week 6).
  Spirometry, used to measure FVC, was performed according to internationally accepted standards. The AUC for FVC was calculated by using the linear trapezoidal rule, based on the changes in FVC from the baseline values, and divided by the observation time (4 hours).
  Definitions:
  AUC=Area under the curve; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); Day 1=Day of the first dose of randomized study drug at Visit 2 (Week 0); FVC=Forced Vital Capacity; FVC AUC(0-4)=Mean FVC after inhalation, measured at prespecified times for up to 4-h observation period (0-4 h), normalized by time;
Time Frame: Baseline, Day 1, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Day 1 | 0.133 [0.087 to 0.179] | 0.192 [0.146 to 0.238] | 0.244 [0.198 to 0.290] | 0.273 [0.227 to 0.319] | 0.036 [-0.010 to 0.082] | 0.311 [0.266 to 0.357]
  Week 6: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  Week 6 | 0.149 [0.089 to 0.210] | 0.203 [0.143 to 0.264] | 0.248 [0.187 to 0.309] | 0.253 [0.194 to 0.313] | 0.000 [-0.062 to 0.061] | 0.353 [0.293 to 0.413]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [0.032 to 0.163]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.156, 95% CI 2-sided [0.091 to 0.221]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.208, 95% CI 2-sided [0.143 to 0.273]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.237, 95% CI 2-sided [0.172 to 0.302]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.276, 95% CI 2-sided [0.211 to 0.341]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 0.076, Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [-0.006 to 0.124]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.046 to 0.176]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [0.075 to 0.205]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; p = 0.116, Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.013 to 0.117]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 0.081, 95% CI 2-sided [0.016 to 0.146]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; p = 0.384, Mixed Models Analysis; Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.036 to 0.094]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 12]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.150, 95% CI 2-sided [0.064 to 0.236]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.204, 95% CI 2-sided [0.118 to 0.290]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.248, 95% CI 2-sided [0.162 to 0.335]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.254, 95% CI 2-sided [0.168 to 0.339]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.354, 95% CI 2-sided [0.268 to 0.439]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.214, Mixed Models Analysis; Mean Difference (Final Values) = 0.054, 95% CI 2-sided [-0.031 to 0.140]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [0.012 to 0.184]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = 0.104, 95% CI 2-sided [0.019 to 0.189]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.313, Mixed Models Analysis; Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.042 to 0.130]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; Week 6 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure. Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.250, Mixed Models Analysis; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [-0.035 to 0.135]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.898, Mixed Models Analysis; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.080 to 0.091]

7. Secondary Outcome: Change From Baseline in FVC Peak(0-4h) on Day 1 and at Week 6
Description: Change from baseline in FVC peak(0-4h) (L) on Day 1 and at the end of treatment at Week 6. Peak FEV1 is defined as the maximum FEV1 observed in the first 4 hours after dose of study medication.
  Definitions:
  Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); Day 1=Day of the first dose of randomized study drug at Visit 2 (Week 0); FVC=Forced Vital Capacity; Peak(0-4h)=Maximum FEV1 between 0 and 4 h.
Time Frame: Baseline, Day 1, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Day 1 | 0.293 [0.241 to 0.345] | 0.372 [0.320 to 0.423] | 0.414 [0.362 to 0.466] | 0.455 [0.403 to 0.506] | 0.213 [0.161 to 0.266] | 0.491 [0.439 to 0.542]
  Week 6: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  Week 6 | 0.322 [0.258 to 0.386] | 0.379 [0.315 to 0.443] | 0.431 [0.366 to 0.495] | 0.427 [0.364 to 0.490] | 0.182 [0.117 to 0.247] | 0.530 [0.467 to 0.594]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Day 1 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed, using linear mixed model for repeated measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [0.006 to 0.153]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.158, 95% CI 2-sided [0.085 to 0.232]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.201, 95% CI 2-sided [0.127 to 0.275]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.241, 95% CI 2-sided [0.168 to 0.315]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.277, 95% CI 2-sided [0.204 to 0.351]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [0.005 to 0.152]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [0.048 to 0.195]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.162, 95% CI 2-sided [0.088 to 0.235]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; p = 0.256, Mixed Models Analysis; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.031 to 0.116]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 10]; Test type: Superiority; p = 0.027, Mixed Models Analysis; Mean Difference (Final Values) = 0.083, 95% CI 2-sided [0.010 to 0.156]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; p = 0.281, Mixed Models Analysis; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.033 to 0.114]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 12]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.141, 95% CI 2-sided [0.050 to 0.232]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.197, 95% CI 2-sided [0.106 to 0.288]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.249, 95% CI 2-sided [0.157 to 0.340]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.245, 95% CI 2-sided [0.155 to 0.336]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.348, 95% CI 2-sided [0.258 to 0.439]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.222, Mixed Models Analysis; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [-0.034 to 0.147]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.020, Mixed Models Analysis; Hazard Ratio, log = 0.108, 95% CI 2-sided [0.017 to 0.199]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [0.015 to 0.195]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.262, Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.039 to 0.143]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.290, Mixed Models Analysis; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.041 to 0.138]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.938, Mixed Models Analysis; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.094 to 0.087]

8. Secondary Outcome: Time to Onset of Action (Change From Baseline in Post-dose FEV1 ≥ 100 mL) on Day 1
Description: Time to onset of action is defined as the time (in minutes) from receiving the study drug on Day 1, until the FEV1 change from baseline is ≥100 mL.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
minutes | 45.1 [34.5 to 66.2] | 32.6 [30.7 to 45.6] | 29.5 [16.3 to 30.8] | 27.3 [16.5 to 30.5] | 240.1 [179.6 to 361.8] | 28.1 [18.0 to 32.1]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using Cox proportional hazards model, including treatment, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and baseline FEV1 value as covariate; Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.21 to 2.24]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.18, 95% CI 2-sided [1.61 to 2.94]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.79, 95% CI 2-sided [2.07 to 3.78]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 3.07, 95% CI 2-sided [2.27 to 4.15]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 3.10, 95% CI 2-sided [2.30 to 4.17]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.052, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.00 to 1.76]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.70, 95% CI 2-sided [1.28 to 2.26]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.87, 95% CI 2-sided [1.41 to 2.48]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.074, Regression, Cox; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.98 to 1.69]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.013, Regression, Cox; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [1.08 to 1.85]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.494, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.84 to 1.44]

9. Secondary Outcome: Number of Patients Achieving Onset of Action - Change From Baseline in Post-dose FEV1 ≥100 mL on Day 1
Description: Number of patients achieving onset of action was defined as a change from baseline in post-dose FEV1 ≥100 mL on Day 1. These are the patients who contributed to the results, reported as median and 95% CI for 'time to onset of action' presented in Outcome Measure 8, above.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Participants | 90 | 103 | 103 | 110 | 74 | 113

10. Secondary Outcome: Change From Baseline in Pre-dose Morning FEV1 at Week 3 and Week 6
Description: Change from baseline in FEV1 at treatment visit 3 (Week 3) and treatment visit 4 (Week 6) of treatment. Spirometry, used to measure FEV1, was performed according to internationally accepted standards.
  Definitions:
  Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose), at Visit 2 (Week 0); FEV1=Forced expiratory volume in the 1st second;
Time Frame: Baseline, Week 3, Week 6
Population: Intention to treat All randomized patients who received at least one dose of the study treatment and with at least one available evaluation of efficacy after baseline (primary or secondary efficacy variables).
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Week 3: number analyzed (Participants) | 121 | 123 | 121 | 123 | 119 | 121
  Week 3 | 0.059 [0.025 to 0.092] | 0.080 [0.047 to 0.114] | 0.122 [0.088 to 0.156] | 0.111 [0.078 to 0.145] | 0.000 [-0.034 to 0.034] | 0.122 [0.089 to 0.156]
  Week 6: number analyzed (Participants) | 117 | 118 | 113 | 122 | 114 | 117
  Week 6 | 0.020 [-0.018 to 0.058] | 0.088 [0.050 to 0.126] | 0.107 [0.068 to 0.145] | 0.130 [0.093 to 0.168] | -0.012 [-0.050 to 0.027] | 0.112 [0.074 to 0.150]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [0.011 to 0.107]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.080, 95% CI 2-sided [0.032 to 0.128]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [0.074 to 0.170]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Hazard Ratio, log = 0.111, 95% CI 2-sided [0.063 to 0.159]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Week 3 Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [0.074 to 0.170]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Week 3 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.377, Mixed Models Analysis; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.026 to 0.069]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Week 3 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [0.015 to 0.111]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Week 3 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.031, Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [0.005 to 0.100]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Week 3 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.085, Mixed Models Analysis; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.006 to 0.089]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Week 3 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.199, Mixed Models Analysis; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.016 to 0.079]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Week 3 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.657, Mixed Models Analysis; Mean Difference (Final Values) = -0.011, 95% CI 2-sided [-0.058 to 0.037]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 12]; Test type: Superiority; p = 0.246, Mixed Models Analysis; Mean Difference (Final Values) = 0.032, 95% CI 2-sided [-0.022 to 0.086]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.100, 95% CI 2-sided [0.046 to 0.154]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.119, 95% CI 2-sided [0.064 to 0.173]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [0.088 to 0.196]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.070 to 0.178]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = 0.068, 95% CI 2-sided [0.014 to 0.121]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.032 to 0.141]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [0.057 to 0.163]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.493, Mixed Models Analysis; Mean Difference (Final Values) = 0.019, 95% CI 2-sided [-0.035 to 0.073]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.119, Mixed Models Analysis; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.011 to 0.096]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.392, Mixed Models Analysis; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.030 to 0.077]

11. Secondary Outcome: Change From Baseline in Pre-Dose Morning Inspiratory Capacity (IC) at Week 3 and Week 6
Description: Change from baseline in IC at treatment Visit 3 (Week 3) and treatment Visit 4 (Week 6). Spirometry was used to measure IC and was performed according to internationally accepted standards.
  Definitions:
  Baseline: value of the measurement recorded at 45 mins pre-dose at Visit 2 (Week 0); IC=Inspiratory capacity;
Time Frame: Baseline, Week 3, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Litres
  Week 3: number analyzed (Participants) | 120 | 122 | 120 | 123 | 118 | 120
  Week 3 | 0.156 [0.090 to 0.222] | 0.137 [0.071 to 0.203] | 0.106 [0.040 to 0.172] | 0.140 [0.074 to 0.205] | 0.047 [-0.020 to 0.113] | 0.090 [0.024 to 0.156]
  Week 6: number analyzed (Participants) | 116 | 117 | 113 | 122 | 113 | 117
  Week 6 | 0.045 [-0.025 to 0.115] | 0.090 [0.021 to 0.160] | 0.136 [0.065 to 0.207] | 0.105 [0.036 to 0.174] | 0.025 [-0.046 to 0.096] | 0.099 [0.029 to 0.169]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model for repeated measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by visit interaction as covariates; Test type: Superiority; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = 0.109, 95% CI 2-sided [0.015 to 0.203]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.058, Mixed Models Analysis; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.003 to 0.184]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.215, Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [-0.035 to 0.153]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 10, analysis 4]; Test type: Superiority; p = 0.051, Mixed Models Analysis; Mean Difference (Final Values) = 0.093, 95% CI 2-sided [-0.001 to 0.187]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.364, Mixed Models Analysis; Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.051 to 0.138]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.694, Mixed Models Analysis; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.112 to 0.074]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.297, Mixed Models Analysis; Mean Difference (Final Values) = -0.050, 95% CI 2-sided [-0.143 to 0.044]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 10, analysis 8]; Test type: Superiority; p = 0.734, Mixed Models Analysis; Mean Difference (Final Values) = -0.016, 95% CI 2-sided [-0.109 to 0.077]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.514, Mixed Models Analysis; Mean Difference (Final Values) = -0.031, 95% CI 2-sided [-0.124 to 0.062]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 10, analysis 10]; Test type: Superiority; p = 0.957, Mixed Models Analysis; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.090 to 0.095]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 10, analysis 11]; Test type: Superiority; p = 0.479, Mixed Models Analysis; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.060 to 0.127]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 12]; Test type: Superiority; p = 0.687, Mixed Models Analysis; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.079 to 0.120]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p = 0.195, Mixed Models Analysis; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [-0.034 to 0.165]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.011 to 0.212]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p = 0.112, Mixed Models Analysis; Mean Difference (Final Values) = 0.080, 95% CI 2-sided [-0.019 to 0.179]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p = 0.147, Mixed Models Analysis; Mean Difference (Final Values) = 0.074, 95% CI 2-sided [-0.026 to 0.174]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.370, Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [-0.054 to 0.144]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.074, Mixed Models Analysis; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [-0.009 to 0.190]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.233, Mixed Models Analysis; Mean Difference (Final Values) = 0.060, 95% CI 2-sided [-0.039 to 0.158]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.369, Mixed Models Analysis; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [-0.054 to 0.145]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.773, Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.084 to 0.112]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.536, Mixed Models Analysis; Mean Difference (Final Values) = -0.031, 95% CI 2-sided [-0.130 to 0.068]

12. Secondary Outcome: Transition Dyspnea Index (TDI) Response (Focal Score ≥1) at Week 3 and Week 6
Description: Number of subjects achieving TDI focal score ≥1, at treatment visit 3 (Week 3) and at treatment visit 4 (Week 6).
  TDI is a validated, interviewer-administered questionnaire that measures changes in dyspnea severity from the baseline established by the BDI questionnaire. TDI consists of the same 24 items and 3 domains as the BDI, with the same 2-week recall period. Each category is rated by 7 grades ranging from -3 (major deterioration) to +3 (major improvement); total score ranging from -9 to +9, with higher scores indicating better outcomes. The minimal clinically important differences (MCID) is considered a change of ≥1 unit. The same investigator or designee interviewed the subject for the BDI and TDI during the study period. A TDI focal score of ≥1 is considered as clinically important.
  Definitions:
  Baseline=The BDI focal score value at Visit 2 (Week 0); BDI=Baseline Dyspnea Index; MCID=Minimal Clinically Important Differences; TDI=Transition Dyspnea Index;
Time Frame: Baseline, Week 3, Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Participants
  Week 3 Focal Score ≥ 1: number analyzed (Participants) | 121 | 123 | 121 | 123 | 119 | 122
  Week 3 Focal Score ≥ 1 | 70 | 78 | 75 | 84 | 67 | 74
  Week 6 Focal Score ≥ 1: number analyzed (Participants) | 118 | 120 | 113 | 122 | 115 | 117
  Week 6 Focal Score ≥ 1 | 74 | 83 | 82 | 91 | 55 | 80
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analysis based on logistic regression model - multiple logistic regression model, with treatment, US regions, smoking status at screening, and BDI as covariates; Test type: Superiority; p = 0.848, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.62 to 1.77]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.264, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.80 to 2.28]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.343, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.76 to 2.18]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 10, analysis 4]; Test type: Superiority; p = 0.042, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.02 to 2.98]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.503, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.71 to 2.02]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.354, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.76 to 2.16]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.447, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.73 to 2.07]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 10, analysis 8]; Test type: Superiority; p = 0.064, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.97 to 2.83]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.867, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.57 to 1.62]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 10, analysis 10]; Test type: Superiority; p = 0.347, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.76 to 2.22]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 10, analysis 11]; Test type: Superiority; p = 0.269, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.79 to 2.32]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; Week 6 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure. Analysis based on logistic regression model - multiple logistic regression model, with treatment, US regions, smoking status at screening, and BDI as covariates; Test type: Superiority; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.12 to 3.30]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.59, 95% CI 2-sided [1.50 to 4.49]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.75 to 5.44]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.42, 95% CI 2-sided [1.94 to 6.02]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.45, 95% CI 2-sided [1.41 to 4.26]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.284, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.78 to 2.35]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.103, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.91 to 2.84]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.045, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.01 to 3.14]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.557, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.67 to 2.12]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.345, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.74 to 2.34]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.732, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.61 to 2.00]

13. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Week 3 and Week 6
Description: Transitional Dyspnea Index (TDI) focal score at treatment visit 3 (Week 3) and treatment visit 4 (Week 6).
  TDI is a validated, interviewer-administered questionnaire that measures changes in dyspnea severity from the baseline established by the BDI questionnaire. TDI consists of the same 24 items and 3 domains as the BDI, with the same 2-week recall period. Each category is rated by 7 grades ranging from -3 (major deterioration) to +3 (major improvement), with a total score ranging from -9 to +9, with higher scores indicating better outcomes. The minimal clinically important differences (MCID) is considered a change of ≥1 unit. The same investigator or designee interviewed the subject for the BDI and TDI during the study period. A TDI focal score of ≥1 is considered as clinically important.
  Definitions:
  Baseline=The BDI focal score value at Visit 2 (Week 0); BDI=Baseline Dyspnea Index; MCID=Minimal Clinically Important Differences; TDI=Transition Dyspnea Index;
Time Frame: Baseline, Week 3, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
score on a scale
  Week 3: number analyzed (Participants) | 121 | 123 | 121 | 123 | 119 | 122
  Week 3 | 1.29 [0.82 to 1.75] | 1.55 [1.09 to 2.01] | 1.54 [1.07 to 2.01] | 1.94 [1.47 to 2.40] | 1.14 [0.67 to 1.61] | 1.66 [1.20 to 2.13]
  Week 6: number analyzed (Participants) | 121 | 123 | 121 | 123 | 119 | 122
  Week 6 | 1.65 [1.18 to 2.11] | 2.02 [1.55 to 2.48] | 2.05 [1.58 to 2.52] | 2.55 [2.09 to 3.01] | 1.03 [0.56 to 1.51] | 2.11 [1.65 to 2.58]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Week 3 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including treatment, visit, treatment by visit interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the BDI, BDI by visit interaction as covariates; Test type: Superiority; p = 0.666, Mixed Models Analysis; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.52 to 0.81]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.224, Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.25 to 1.07]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.239, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.27 to 1.06]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 10, analysis 4]; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [0.13 to 1.46]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.124, Mixed Models Analysis; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.14 to 1.19]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.432, Mixed Models Analysis; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.39 to 0.92]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.454, Mixed Models Analysis; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.41 to 0.91]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 10, analysis 8]; Test type: Superiority; p = 0.053, Mixed Models Analysis; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-0.01 to 1.31]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.973, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.67 to 0.65]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 10, analysis 10]; Test type: Superiority; p = 0.247, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.27 to 1.04]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 10, analysis 11]; Test type: Superiority; p = 0.235, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.26 to 1.06]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 4, analysis 12]; Test type: Superiority; p = 0.071, Mixed Models Analysis; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.05 to 1.28]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [0.32 to 1.64]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 3, analysis 14]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [0.35 to 1.68]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [0.86 to 2.18]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 3, analysis 16]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.41 to 1.75]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.271, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.29 to 1.03]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 3, analysis 18]; Test type: Superiority; p = 0.235, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.26 to 1.06]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.25 to 1.56]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 3, analysis 20]; Test type: Superiority; p = 0.923, Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.63 to 0.69]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.108, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.12 to 1.19]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 3, analysis 22]; Test type: Superiority; p = 0.134, Mixed Models Analysis; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.16 to 1.16]

14. Secondary Outcome: Change From Baseline in Percentage of Rescue Medication-Free Days During Inter-Visit Periods and the Entire Treatment Period
Description: Evaluate the number of rescue medication-free days compared with baseline. Results are shown as percentage (%) of rescue medication-free days; an increased value indicates improvement from baseline.
  Definitions:
  Baseline=Data recorded during the run-in period (a 2-week period prior to randomization to study treatment and study drug intake); Inter-visit period 1=Starts at randomization to treatment (Visit 2, Week 0) and runs to the day before the subject returns to the clinic (Visit 3, Week 3); Inter-visit period 2=Starts when the subject returns to the clinic (Visit 3, Week 3) and runs to the end of the randomized treatment period (Visit 4, Week 6); Entire Treatment period=From day of randomization to drug intake to the end of the randomized treatment period (Visit 4, Week 6); Randomization=Randomization to study drug treatment (Visit 2, Week 0).
Time Frame: Baseline, Inter-visit period 1, Inter-visit period 2, Entire treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: % of of rescue medication-free days
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
% of of rescue medication-free days
  Inter-visit period 1: number analyzed (Participants) | 111 | 114 | 112 | 113 | 111 | 102
  Inter-visit period 1 | 16.78 [12.02 to 21.54] | 15.67 [10.96 to 20.39] | 15.55 [10.79 to 20.31] | 18.19 [13.44 to 22.94] | 8.90 [4.12 to 13.68] | 13.51 [8.52 to 18.50]
  Inter-visit period 2: number analyzed (Participants) | 109 | 110 | 103 | 113 | 105 | 97
  Inter-visit period 2 | 13.83 [8.69 to 18.97] | 15.51 [10.40 to 20.62] | 14.03 [8.83 to 19.23] | 18.15 [13.04 to 23.27] | 7.07 [1.87 to 12.27] | 11.27 [5.85 to 16.69]
  Entire treatment period: number analyzed (Participants) | 108 | 110 | 103 | 113 | 105 | 97
  Entire treatment period | 15.30 [10.61 to 20.00] | 15.59 [10.93 to 20.25] | 14.79 [10.07 to 19.50] | 18.17 [13.49 to 22.86] | 7.98 [3.25 to 12.72] | 12.39 [7.45 to 17.32]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including inter-visit period, treatment by inter-visit period interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by inter-visit period interaction as covariates; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Final Values) = 7.88, 95% CI 2-sided [1.13 to 14.63]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.048, Mixed Models Analysis; Mean Difference (Final Values) = 6.78, 95% CI 2-sided [0.07 to 13.48]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.053, Mixed Models Analysis; Mean Difference (Final Values) = 6.65, 95% CI 2-sided [-0.09 to 13.40]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 9.29, 95% CI 2-sided [2.55 to 16.04]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.191, Mixed Models Analysis; Mean Difference (Final Values) = 4.61, 95% CI 2-sided [-2.31 to 11.53]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.747, Mixed Models Analysis; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-7.80 to 5.60]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.720, Mixed Models Analysis; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-7.96 to 5.50]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.680, Mixed Models Analysis; Mean Difference (Final Values) = 1.41, 95% CI 2-sided [-5.31 to 8.14]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.971, Mixed Models Analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-6.82 to 6.57]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.460, Mixed Models Analysis; Mean Difference (Final Values) = 2.52, 95% CI 2-sided [-4.17 to 9.21]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Inter-Visit period 1 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.441, Mixed Models Analysis; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [-4.09 to 9.37]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.070, Mixed Models Analysis; Mean Difference (Final Values) = 6.76, 95% CI 2-sided [-0.55 to 14.08]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = 8.44, 95% CI 2-sided [1.16 to 15.72]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.064, Mixed Models Analysis; Mean Difference (Final Values) = 6.96, 95% CI 2-sided [-0.40 to 14.31]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 11.08, 95% CI 2-sided [3.79 to 18.38]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.274, Mixed Models Analysis; Mean Difference (Final Values) = 4.20, 95% CI 2-sided [-3.32 to 11.72]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.649, Mixed Models Analysis; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-5.57 to 8.93]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.958, Mixed Models Analysis; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-7.12 to 7.51]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.242, Mixed Models Analysis; Mean Difference (Final Values) = 4.32, 95% CI 2-sided [-2.93 to 11.58]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.690, Mixed Models Analysis; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-8.77 to 5.81]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.473, Mixed Models Analysis; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [-4.58 to 9.87]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; Inter-Visit period 2 Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.267, Mixed Models Analysis; Mean Difference (Final Values) = 4.13, 95% CI 2-sided [-3.17 to 11.43]
Statistical Analysis 23: Comparison: Treatment A vs Treatment E; Entire treatment period Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.032, Mixed Models Analysis; Mean Difference (Final Values) = 7.32, 95% CI 2-sided [0.65 to 13.99]
Statistical Analysis 24: Comparison: Treatment B vs Treatment E; Entire treatment period Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Final Values) = 7.61, 95% CI 2-sided [0.97 to 14.24]
Statistical Analysis 25: Comparison: Treatment C vs Treatment E; Entire treatment period Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.046, Mixed Models Analysis; Mean Difference (Final Values) = 6.80, 95% CI 2-sided [0.12 to 13.49]
Statistical Analysis 26: Comparison: Treatment D vs Treatment E; Entire treatment period Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 10.19, 95% CI 2-sided [3.52 to 16.85]
Statistical Analysis 27: Comparison: Treatment E vs Treatment F; Entire treatment period Comparison treatment groups for this analysis were: Treatment F (Tiotropium 18 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.207, Mixed Models Analysis; Mean Difference (Final Values) = 4.40, 95% CI 2-sided [-2.45 to 11.25]
Statistical Analysis 28: Comparison: Treatment A vs Treatment B; Entire treatment period Comparison treatment groups for this analysis were: Treatment B (CHF 5259 pMDI 25 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.932, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-6.33 to 6.91]
Statistical Analysis 29: Comparison: Treatment A vs Treatment C; Entire treatment period Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.879, Mixed Models Analysis; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-7.17 to 6.14]
Statistical Analysis 30: Comparison: Treatment A vs Treatment D; Entire treatment period Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment A (CHF 5259 pMDI 12.5 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.396, Mixed Models Analysis; Mean Difference (Final Values) = 2.87, 95% CI 2-sided [-3.77 to 9.50]
Statistical Analysis 31: Comparison: Treatment B vs Treatment C; Entire treatment period Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.812, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-7.44 to 5.83]
Statistical Analysis 32: Comparison: Treatment B vs Treatment D; Entire treatment period Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.444, Mixed Models Analysis; Mean Difference (Final Values) = 2.58, 95% CI 2-sided [-4.03 to 9.19]
Statistical Analysis 33: Comparison: Treatment C vs Treatment D; Entire treatment period Comparison treatment groups for this analysis were: Treatment D (CHF 5259 pMDI 100 μg TDD) versus Treatment C (CHF 5259 pMDI 50 μg TDD). Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.319, Mixed Models Analysis; Mean Difference (Final Values) = 3.38, 95% CI 2-sided [-3.27 to 10.04]

15. Secondary Outcome: Change From Baseline in Average Use of Rescue Medication During Inter-Visit Periods and the Entire Treatment Period
Description: Evaluate the change from baseline in average use of rescue medication (number of puffs/day) during the inter-visit periods and the entire treatment period.
  Results are shown as number of puffs/day; a decrease (implies improvement) from baseline in average use of rescue medication.
  Definitions:
  Baseline=Data recorded during the run-in period (a 2-week period prior to randomization to study treatment and study drug intake); Inter-visit period 1=Starts at randomization to treatment (Visit 2, Week 0) and runs to the day before the subject returns to the clinic (Visit 3 (Week 3); Inter-visit period 2=Starts when the subject returns to the clinic (Visit 3, Week 3) and runs to the end of the randomized treatment period (Visit 4, Week 6); Entire Treatment period=From day of randomization to drug intake to the end of the randomized treatment period (Visit 4, Week 6); Randomization=Randomization to study drug treatment (Visit 2, Week 0);
Time Frame: Baseline, Inter-visit period 1, Inter-visit period 2, Entire treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of puffs/day
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Number of puffs/day
  Inter-visit period 1: number analyzed (Participants) | 111 | 114 | 112 | 113 | 111 | 102
  Inter-visit period 1 | -0.72 [-0.90 to -0.55] | -0.58 [-0.75 to -0.41] | -0.53 [-0.70 to -0.35] | -0.71 [-0.89 to -0.54] | -0.30 [-0.47 to -0.12] | -0.52 [-0.70 to -0.34]
  Inter-visit period 2: number analyzed (Participants) | 109 | 110 | 103 | 113 | 105 | 97
  Inter-visit period 2 | -0.59 [-0.78 to -0.39] | -0.50 [-0.69 to -0.30] | -0.51 [-0.71 to -0.31] | -0.69 [-0.89 to -0.50] | -0.17 [-0.37 to 0.03] | -0.40 [-0.61 to -0.19]
  Entire treatment period: number analyzed (Participants) | 108 | 110 | 103 | 113 | 105 | 97
  Entire treatment period | -0.66 [-0.83 to -0.48] | -0.54 [-0.71 to -0.37] | -0.52 [-0.70 to -0.34] | -0.70 [-0.88 to -0.53] | -0.23 [-0.41 to -0.06] | -0.46 [-0.64 to -0.28]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Inter-visit period 1 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed, using linear mixed model repeated for measurements (MMRM), including treatment, inter-visit period, treatment by inter-visit period interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by inter-visit period interaction as covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.67 to -0.18]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.53 to -0.04]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.067, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.47 to 0.02]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.66 to -0.17]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.084, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.47 to 0.03]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.243, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.10 to 0.39]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p = 0.112, Mixed Models Analysis; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.05 to 0.44]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 14, analysis 8]; Test type: Superiority; p = 0.929, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.23 to 0.26]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p = 0.668, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.19 to 0.30]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 14, analysis 10]; Test type: Superiority; p = 0.281, Mixed Models Analysis; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.38 to 0.11]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 14, analysis 11]; Test type: Superiority; p = 0.134, Mixed Models Analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.43 to 0.06]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 14, analysis 12]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.70 to -0.14]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 14, analysis 13]; Test type: Superiority; p = 0.020, Mixed Models Analysis; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.61 to -0.05]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 14, analysis 14]; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.62 to -0.06]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 14, analysis 15]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.80 to -0.24]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 14, analysis 16]; Test type: Superiority; p = 0.115, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.52 to 0.06]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 14, analysis 17]; Test type: Superiority; p = 0.532, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.19 to 0.36]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 14, analysis 18]; Test type: Superiority; p = 0.603, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.21 to 0.35]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 14, analysis 19]; Test type: Superiority; p = 0.460, Mixed Models Analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.38 to 0.17]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; Inter-visit period 2 Comparison treatment groups for this analysis were: Treatment C (CHF 5259 pMDI 50 μg TDD) versus Treatment B (CHF 5259 pMDI 25 μg TDD. Statistical analysis was performed as described for the statistical analysis 1 of this outcome measure; Test type: Superiority; p = 0.921, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.29 to 0.26]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 14, analysis 21]; Test type: Superiority; p = 0.172, Mixed Models Analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.47 to 0.08]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 14, analysis 22]; Test type: Superiority; p = 0.210, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.46 to 0.10]
Statistical Analysis 23: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 14, analysis 23]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.67 to -0.17]
Statistical Analysis 24: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 14, analysis 24]; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.55 to -0.06]
Statistical Analysis 25: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 14, analysis 25]; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.54 to -0.04]
Statistical Analysis 26: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 14, analysis 26]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.72 to -0.22]
Statistical Analysis 27: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 14, analysis 27]; Test type: Superiority; p = 0.083, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.48 to 0.03]
Statistical Analysis 28: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 14, analysis 28]; Test type: Superiority; p = 0.355, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.13 to 0.36]
Statistical Analysis 29: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 14, analysis 29]; Test type: Superiority; p = 0.283, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.11 to 0.38]
Statistical Analysis 30: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 14, analysis 30]; Test type: Superiority; p = 0.712, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.29 to 0.20]
Statistical Analysis 31: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority; p = 0.877, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.23 to 0.27]
Statistical Analysis 32: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 14, analysis 32]; Test type: Superiority; p = 0.195, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.41 to 0.08]
Statistical Analysis 33: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 14, analysis 33]; Test type: Superiority; p = 0.150, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.43 to 0.07]

16. Secondary Outcome: Change From Baseline in Average EXACT-Respiratory Symptom (E-RS) Total Score During Inter-Visit Periods and the Entire Treatment Period
Description: Change from baseline in average EXACT-Respiratory Symptom (E-RS) total score during inter-visit periods and the entire treatment period
  E-RS in COPD uses 11 respiratory symptom items from the 14-item EXAcerbations of COPD tool (EXACT). E-RS total score quantifies respiratory symptom severity on a scale ranging from 0 to 40. Higher E-RS total scores indicate more severe symptoms and a declining total score indicates health improvement. E-RS questionnaire was completed by the patient each evening (e-diary).
  Definitions:
  For details on baseline, inter-visit periods, and the entire treatment period, please refer to outcome measure #15.
Time Frame: Baseline, Inter-visit period 1, Inter-visit period 2, Entire treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
score on a scale
  Inter-visit period 1: number analyzed (Participants) | 111 | 114 | 112 | 113 | 111 | 102
  Inter-visit period 1 | -1.681 [-2.236 to -1.127] | -1.539 [-2.087 to -0.990] | -1.941 [-2.495 to -1.388] | -1.663 [-2.215 to -1.111] | -0.714 [-1.272 to -0.157] | -1.280 [-1.862 to -0.698]
  Inter-visit period 2: number analyzed (Participants) | 109 | 110 | 103 | 112 | 105 | 97
  Inter-visit period 2 | -2.030 [-2.694 to -1.365] | -1.840 [-2.499 to -1.180] | -2.147 [-2.818 to -1.475] | -2.077 [-2.737 to -1.417] | -0.681 [-1.353 to -0.009] | -1.505 [-2.206 to -0.803]
  Entire treatment period: number analyzed (Participants) | 108 | 110 | 103 | 112 | 105 | 97
  Entire treatment period | -1.855 [-2.433 to -1.278] | -1.689 [-2.262 to -1.116] | -2.044 [-2.624 to -1.464] | -1.870 [-2.445 to -1.295] | -0.698 [-1.280 to -0.115] | -1.393 [-2.001 to -0.784]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Inter-visit period 1 Comparison treatment groups for this analysis were: Treatment A (CHF 5259 pMDI 12.5 μg TDD) versus Treatment E (Placebo). Analyzed using linear mixed model repeated for measurements (MMRM), including treatment, inter-visit period, treatment by inter-visit period interaction, US regions (Midwest, Northeast, South and West), and smoking status at screening as fixed effects, and the baseline value, and baseline by inter-visit period interaction as covariates; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -0.967, 95% CI 2-sided [-1.753 to -0.181]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.039, Mixed Models Analysis; Mean Difference (Final Values) = -0.824, 95% CI 2-sided [-1.606 to -0.043]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -1.227, 95% CI 2-sided [-2.012 to -0.441]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.018, Mixed Models Analysis; Mean Difference (Final Values) = -0.949, 95% CI 2-sided [-1.733 to -0.164]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 14, analysis 5]; Test type: Superiority; p = 0.169, Mixed Models Analysis; Mean Difference (Final Values) = -0.566, 95% CI 2-sided [-1.374 to 0.242]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.720, Mixed Models Analysis; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [-0.638 to 0.923]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 14, analysis 7]; Test type: Superiority; p = 0.515, Mixed Models Analysis; Mean Difference (Final Values) = -0.260, 95% CI 2-sided [-1.043 to 0.523]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 14, analysis 8]; Test type: Superiority; p = 0.963, Mixed Models Analysis; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.764 to 0.800]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 14, analysis 9]; Test type: Superiority; p = 0.311, Mixed Models Analysis; Mean Difference (Final Values) = -0.402, 95% CI 2-sided [-1.182 to 0.377]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 14, analysis 10]; Test type: Superiority; p = 0.754, Mixed Models Analysis; Mean Difference (Final Values) = -0.124, 95% CI 2-sided [-0.903 to 0.654]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 14, analysis 11]; Test type: Superiority; p = 0.485, Mixed Models Analysis; Mean Difference (Final Values) = 0.278, 95% CI 2-sided [-0.503 to 1.060]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 14, analysis 12]; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -1.349, 95% CI 2-sided [-2.294 to -0.403]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 14, analysis 13]; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -1.159, 95% CI 2-sided [-2.100 to -0.218]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 14, analysis 14]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -1.466, 95% CI 2-sided [-2.416 to -0.516]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 14, analysis 15]; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1.396, 95% CI 2-sided [-2.337 to -0.454]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 14, analysis 16]; Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Final Values) = -0.824, 95% CI 2-sided [-1.797 to 0.150]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 14, analysis 17]; Test type: Superiority; p = 0.690, Mixed Models Analysis; Mean Difference (Final Values) = 0.190, 95% CI 2-sided [-0.746 to 1.126]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 14, analysis 18]; Test type: Superiority; p = 0.808, Mixed Models Analysis; Mean Difference (Final Values) = -0.117, 95% CI 2-sided [-1.061 to 0.827]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 14, analysis 19]; Test type: Superiority; p = 0.922, Mixed Models Analysis; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.983 to 0.889]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 14, analysis 20]; Test type: Superiority; p = 0.522, Mixed Models Analysis; Mean Difference (Final Values) = -0.307, 95% CI 2-sided [-1.248 to 0.634]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 14, analysis 21]; Test type: Superiority; p = 0.618, Mixed Models Analysis; Mean Difference (Final Values) = -0.237, 95% CI 2-sided [-1.170 to 0.696]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 14, analysis 22]; Test type: Superiority; p = 0.884, Mixed Models Analysis; Mean Difference (Final Values) = 0.070, 95% CI 2-sided [-0.871 to 1.012]
Statistical Analysis 23: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 14, analysis 23]; Test type: Superiority; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -1.158, 95% CI 2-sided [-1.978 to -0.337]
Statistical Analysis 24: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 14, analysis 24]; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = -0.992, 95% CI 2-sided [-1.808 to -0.175]
Statistical Analysis 25: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 14, analysis 25]; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.346, 95% CI 2-sided [-2.168 to -0.524]
Statistical Analysis 26: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 14, analysis 26]; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -1.172, 95% CI 2-sided [-1.991 to -0.353]
Statistical Analysis 27: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 14, analysis 27]; Test type: Superiority; p = 0.107, Mixed Models Analysis; Mean Difference (Final Values) = -0.695, 95% CI 2-sided [-1.539 to 0.149]
Statistical Analysis 28: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 14, analysis 28]; Test type: Superiority; p = 0.689, Mixed Models Analysis; Mean Difference (Final Values) = 0.166, 95% CI 2-sided [-0.648 to 0.980]
Statistical Analysis 29: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 14, analysis 29]; Test type: Superiority; p = 0.651, Mixed Models Analysis; Mean Difference (Final Values) = -0.188, 95% CI 2-sided [-1.007 to 0.630]
Statistical Analysis 30: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 14, analysis 30]; Test type: Superiority; p = 0.973, Mixed Models Analysis; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-0.830 to 0.801]
Statistical Analysis 31: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 14, analysis 31]; Test type: Superiority; p = 0.393, Mixed Models Analysis; Mean Difference (Final Values) = -0.355, 95% CI 2-sided [-1.170 to 0.461]
Statistical Analysis 32: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 14, analysis 32]; Test type: Superiority; p = 0.663, Mixed Models Analysis; Mean Difference (Final Values) = -0.181, 95% CI 2-sided [-0.993 to 0.632]
Statistical Analysis 33: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 14, analysis 33]; Test type: Superiority; p = 0.676, Mixed Models Analysis; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [-0.643 to 0.991]

17. Secondary Outcome: Vital Signs -- Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP)
Description: Vital signs -- Systolic blood pressure (SBP), Diastolic blood pressure (DBP) were measured at prespecified times, using a 12-Lead single ECGs were recorded at all study visits (pre-dose at V1 (Week -2) and V3 (Week 3), as well as at pre-dose and 1.5 hours post-dose at Visit 2 (Week 0) and Visit 4 (Week 6).
  Results are shown by treatment group, as change from baseline (in mmHg) for representative timepoints.
  Definitions:
  Baseline=Values recorded pre-dose (Visit 2, Week 0); Day 1=Day of the first dose of randomized study drug (Visit 2, Week 0);
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
mmHg
  SBP, Day 1, 30 min post dose: number analyzed (Participants) | 121 | 122 | 121 | 123 | 121 | 122
  SBP, Day 1, 30 min post dose | -1.4 [-31 to 25] | -0.4 [-24 to 24] | -2.0 [-31 to 24] | -1.9 [-32 to 34] | -0.9 [-25 to 26] | -1.2 [-32 to 30]
  DBP, Day 1, 30 min post dose: number analyzed (Participants) | 121 | 122 | 121 | 123 | 121 | 122
  DBP, Day 1, 30 min post dose | -0.7 [-21 to 14] | -0.6 [-15 to 15] | -2.1 [-20 to 11] | -1.4 [-28 to 17] | -0.8 [-15 to 12] | 0.1 [-27 to 22]
  SBP, Day 1, 1,5 h post dose | 0.3 [-33 to 24] | -1.1 [-29 to 36] | -0.6 [-33 to 24] | -1.8 [-34 to 22] | 0.2 [-25 to 33] | -1.5 [-30 to 34]
  DBP, Day 1, 1,5 h post dose | -0.7 [-20 to 17] | -1.8 [-22 to 20] | -1.7 [-23 to 13] | -1.6 [-31 to 17] | -1.7 [-18 to 14] | -1.5 [-23 to 23]
  SBP, Day 1, 11 h post dose: number analyzed (Participants) | 121 | 123 | 121 | 122 | 121 | 123
  SBP, Day 1, 11 h post dose | 1.1 [-27 to 34] | 2.0 [-25 to 39] | -0.0 [-34 to 34] | 1.7 [-26 to 39] | 1.9 [-35 to 56] | 0.9 [-25 to 48]
  DBP, Day 1, 11 h post dose: number analyzed (Participants) | 121 | 123 | 121 | 122 | 121 | 123
  DBP, Day 1, 11 h post dose | -0.9 [-20 to 17] | 0.3 [-18 to 21] | -1.6 [-27 to 17] | -1.4 [-18 to 20] | -1.0 [-25 to 22] | -1.2 [-19 to 27]
  SBP, Week 6, pre-dose: number analyzed (Participants) | 117 | 119 | 113 | 122 | 114 | 117
  SBP, Week 6, pre-dose | 0.4 [-34 to 31] | 0.8 [-50 to 34] | 0.4 [-27 to 47] | -1.0 [-36 to 47] | 1.6 [-32 to 46] | 1.3 [-33 to 63]
  DBP, Week 6, pre-dose: number analyzed (Participants) | 117 | 119 | 113 | 122 | 114 | 117
  DBP, Week 6, pre-dose | 0.4 [-32 to 25] | 0.5 [-23 to 21] | -0.3 [-16 to 18] | -1.0 [-28 to 25] | 0.0 [-26 to 18] | -0.2 [-30 to 20]
  SBP, Week 6, 30 min post dose: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  SBP, Week 6, 30 min post dose | -1.6 [-35 to 27] | -0.9 [-62 to 39] | -0.5 [-34 to 42] | -2.5 [-41 to 35] | 0.5 [-30 to 42] | 0.1 [-35 to 54]
  DBP, Week 6, 30 min post dose: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  DBP, Week 6, 30 min post dose | -0.7 [-24 to 21] | -0.9 [-28 to 19] | -1.5 [-24 to 19] | -2.0 [-25 to 22] | -0.8 [-24 to 24] | -1.2 [-26 to 24]
  SBP, Week 6, 1,5 h post dose: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  SBP, Week 6, 1,5 h post dose | -1.3 [-32 to 31] | -0.6 [-31 to 36] | -0.5 [-34 to 47] | -2.3 [-42 to 40] | 0.1 [-34 to 49] | 0.5 [-34 to 67]
  DBP, Week 6, 1,5 h post dose: number analyzed (Participants) | 114 | 113 | 110 | 120 | 110 | 116
  DBP, Week 6, 1,5 h post dose | -1.0 [-28 to 21] | -2.7 [-28 to 16] | -2.0 [-21 to 17] | -2.3 [-30 to 22] | -1.1 [-31 to 19] | -0.6 [-28 to 33]
  SBP, Week 6, 11 h post dose: number analyzed (Participants) | 113 | 112 | 109 | 118 | 109 | 114
  SBP, Week 6, 11 h post dose | 0.2 [-38 to 36] | 1.5 [-26 to 36] | 0.5 [-31 to 53] | 2.2 [-37 to 53] | 3.2 [-25 to 66] | 2.0 [-26 to 45]
  DBP, Week 6, 11 h post dose: number analyzed (Participants) | 113 | 112 | 109 | 118 | 109 | 114
  DBP, Week 6, 11 h post dose | -0.9 [-24 to 21] | -2.0 [-27 to 19] | -2.3 [-25 to 25] | -1.4 [-27 to 21] | -1.0 [-27 to 20] | -0.7 [-17 to 21]

18. Secondary Outcome: Change From Baseline in 24-Hour Holter Electrocardiogram (ECG) Parameters - Heart Rate (HR)
Description: Change from baseline in 24-Hour Holter electrocardiogram (ECG) parameters - Heart rate (HR)
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5m, +55m, and at +2.5 h.
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
bpm
  HR, Day 1, 5 min post dose: number analyzed (Participants) | 88 | 88 | 94 | 85 | 95 | 90
  HR, Day 1, 5 min post dose | -8.85 [-57.3 to 16.3] | -6.62 [-53.7 to 22.3] | -7.78 [-44.0 to 14.3] | -7.64 [-41.3 to 19.0] | -4.84 [-39.7 to 31.7] | -5.54 [-34.3 to 24.3]
  HR, Day 1, 55 min post dose: number analyzed (Participants) | 94 | 95 | 100 | 93 | 103 | 96
  HR, Day 1, 55 min post dose | -7.19 [-45.7 to 12.0] | -8.29 [-33.3 to 10.3] | -8.28 [-40.0 to 27.7] | -9.59 [-74.0 to 17.3] | -7.44 [-49.3 to 36.3] | -7.19 [-41.3 to 37.7]
  HR, Day 1, 2.5 h post dose: number analyzed (Participants) | 102 | 103 | 102 | 101 | 105 | 105
  HR, Day 1, 2.5 h post dose | -7.57 [-51.7 to 19.3] | -6.75 [-51.0 to 16.7] | -9.20 [-46.7 to 26.7] | -7.46 [-94.7 to 21.0] | -6.12 [-45.7 to 30.3] | -8.96 [-40.0 to 18.0]
  HR, Day before Week 6, 5 min post dose: number analyzed (Participants) | 82 | 78 | 75 | 80 | 83 | 84
  HR, Day before Week 6, 5 min post dose | -1.72 [-56.3 to 34.3] | -1.06 [-47.0 to 44.3] | -1.61 [-37.0 to 30.3] | -1.85 [-31.3 to 36.0] | 3.92 [-31.3 to 47.0] | 1.70 [-28.7 to 25.7]
  HR, Day before Week 6, 55 min post dose: number analyzed (Participants) | 95 | 91 | 89 | 91 | 92 | 93
  HR, Day before Week 6, 55 min post dose | -1.52 [-40.7 to 33.0] | 0.41 [-30.0 to 33.0] | -1.10 [-37.3 to 49.3] | -1.40 [-77.7 to 25.0] | 1.12 [-41.3 to 44.2] | 1.22 [-25.3 to 36.7]
  HR, Day before Week 6, 2.5 h post dose: number analyzed (Participants) | 98 | 99 | 93 | 99 | 92 | 100
  HR, Day before Week 6, 2.5 h post dose | -2.30 [-48.0 to 22.3] | -0.01 [-58.3 to 44.3] | -1.13 [-39.3 to 26.3] | -0.73 [-42.0 to 39.7] | 2.49 [-35.7 to 43.7] | -1.47 [-34.7 to 44.0]

19. Secondary Outcome: Change From Baseline in 24-Hour Holter Electrocardiogram (ECG) Parameters - PR Interval
Description: Change from baseline in 24-Hour Holter electrocardiogram (ECG) parameters - PR Interval
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values were recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5 min, +55 min, and at +2.5 h.
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
msec
  PR Interval, Day 1, 5 min post dose: number analyzed (Participants) | 84 | 85 | 93 | 85 | 94 | 88
  PR Interval, Day 1, 5 min post dose | 7.24 [-23.0 to 54.7] | 6.53 [-17.3 to 48.3] | 6.08 [-36.0 to 37.3] | 6.71 [-14.3 to 41.7] | 3.06 [-20.7 to 33.7] | 4.90 [-18.3 to 30.7]
  PR Interval, Day 1, 55 min post dose: number analyzed (Participants) | 89 | 92 | 98 | 93 | 101 | 94
  PR Interval, Day 1, 55 min post dose | 7.20 [-23.0 to 59.7] | 6.89 [-24.3 to 120.7] | 8.21 [-26.7 to 42.3] | 6.77 [-20.0 to 49.3] | 4.38 [-35.7 to 36.0] | 4.77 [-32.7 to 40.0]
  PR Interval, Day 1, 2.5 h post dose: number analyzed (Participants) | 96 | 100 | 98 | 101 | 103 | 104
  PR Interval, Day 1, 2.5 h post dose | 8.48 [-20.3 to 77.7] | 9.38 [-37.0 to 131.3] | 7.58 [-18.7 to 91.3] | 6.16 [-22.0 to 47.3] | 5.84 [-27.0 to 38.7] | 4.25 [-36.7 to 40.7]
  PR Interval, Day before Week 6, 5 min post dose: number analyzed (Participants) | 77 | 76 | 74 | 79 | 82 | 82
  PR Interval, Day before Week 6, 5 min post dose | 0.44 [-27.7 to 39.3] | 1.36 [-30.0 to 59.0] | -0.11 [-54.3 to 26.7] | 3.88 [-33.3 to 204.0] | -1.36 [-48.3 to 31.7] | 0.82 [-23.3 to 37.2]
  PR Interval, Day before Week 6, 55 min post dose: number analyzed (Participants) | 90 | 89 | 87 | 90 | 90 | 91
  PR Interval, Day before Week 6, 55 min post dose | 0.88 [-47.3 to 32.3] | 2.37 [-53.7 to 38.7] | 1.91 [-76.3 to 37.7] | 0.82 [-33.3 to 50.0] | -1.13 [-46.0 to 48.3] | -1.66 [-48.0 to 25.0]
  PR Interval, Day before Week 6, 2.5 h post dose: number analyzed (Participants) | 92 | 97 | 89 | 98 | 90 | 99
  PR Interval, Day before Week 6, 2.5 h post dose | 2.50 [-38.7 to 40.0] | 3.01 [-54.7 to 76.0] | 0.16 [-59.0 to 81.0] | 0.84 [-30.0 to 61.7] | -1.22 [-59.0 to 47.7] | -1.94 [-47.0 to 55.3]

20. Secondary Outcome: Change From Baseline in 24-Hour Holter Electrocardiogram (ECG) Parameters - QRS Interval
Description: Change from baseline in 24-Hour Holter electrocardiogram (ECG) parameters - QRS Interval
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values were recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5 min, +55 min, and at +2.5 h.
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
msec
  QRS Interval, Day 1, 5 min post dose: number analyzed (Participants) | 88 | 88 | 94 | 84 | 95 | 90
  QRS Interval, Day 1, 5 min post dose | 1.18 [-15.0 to 14.7] | 0.05 [-17.7 to 16.7] | 1.50 [-12.0 to 17.7] | 1.99 [-6.0 to 16.7] | 0.45 [-13.0 to 20.3] | 1.50 [-14.0 to 13.0]
  QRS Interval, Day 1, 55 min post dose: number analyzed (Participants) | 94 | 95 | 99 | 93 | 103 | 96
  QRS Interval, Day 1, 55 min post dose | 0.97 [-16.3 to 15.0] | 1.19 [-18.0 to 31.0] | 1.21 [-14.7 to 20.0] | 1.56 [-11.0 to 14.7] | 0.14 [-13.7 to 13.7] | 1.70 [-13.3 to 16.3]
  QRS Interval, Day 1, 2.5 h post dose: number analyzed (Participants) | 102 | 103 | 100 | 100 | 105 | 105
  QRS Interval, Day 1, 2.5 h post dose | 1.38 [-14.0 to 15.0] | 2.40 [-15.3 to 23.7] | 1.80 [-23.0 to 17.3] | 1.50 [-17.8 to 27.3] | 0.64 [-10.3 to 20.8] | 0.86 [-20.7 to 18.7]
  QRS Interval, Day before Week 6, 5 min post dose: number analyzed (Participants) | 82 | 78 | 75 | 79 | 83 | 84
  QRS Interval, Day before Week 6, 5 min post dose | 0.61 [-23.3 to 34.0] | -1.76 [-76.0 to 17.3] | 0.43 [-15.0 to 13.3] | 2.00 [-8.7 to 67.3] | 0.45 [-22.3 to 44.3] | 0.69 [-17.0 to 17.5]
  QRS Interval, Day before Week 6, 55 min post dose: number analyzed (Participants) | 95 | 91 | 88 | 91 | 92 | 93
  QRS Interval, Day before Week 6, 55 min post dose | 1.12 [-10.7 to 29.3] | -0.09 [-76.7 to 30.0] | 0.85 [-18.3 to 13.7] | 2.38 [-10.7 to 62.3] | 0.77 [-16.0 to 53.7] | 0.42 [-20.3 to 17.7]
  QRS Interval, Day before Week 6, 2.5 h post dose: number analyzed (Participants) | 98 | 99 | 92 | 98 | 92 | 100
  QRS Interval, Day before Week 6, 2.5 h post dose | 1.49 [-14.0 to 40.0] | 0.74 [-73.0 to 25.0] | 0.30 [-18.3 to 24.0] | 2.18 [-18.2 to 59.3] | 1.14 [-14.7 to 43.7] | 1.35 [-15.7 to 27.0]

21. Secondary Outcome: Change From Baseline in 24-Hour Holter Electrocardiogram (ECG) Parameters - Fridericia-corrected QT Interval (QTcF)
Description: Change from baseline in 24-Hour Holter electrocardiogram (ECG) parameters - Fridericia-corrected QT interval (QTcF).
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5 min, +55 min, and at +2.5 h.
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
msec
  QTcF, Day 1, 5 min post dose: number analyzed (Participants) | 88 | 88 | 94 | 84 | 95 | 90
  QTcF, Day 1, 5 min post dose | 3.62 [-38.0 to 39.7] | 5.37 [-48.7 to 55.7] | 6.81 [-34.0 to 39.7] | 6.25 [-30.3 to 52.7] | 3.59 [-33.3 to 50.3] | 5.56 [-21.7 to 53.3]
  QTcF, Day 1, 55 min post dose: number analyzed (Participants) | 94 | 95 | 98 | 93 | 103 | 96
  QTcF, Day 1, 55 min post dose | 8.37 [-35.3 to 47.0] | 5.41 [-52.3 to 45.0] | 6.72 [-43.7 to 40.7] | 9.90 [-20.3 to 67.7] | 6.04 [-34.7 to 61.3] | 5.43 [-24.7 to 42.5]
  QTcF, Day 1, 2.5 h post dose: number analyzed (Participants) | 101 | 103 | 98 | 100 | 105 | 105
  QTcF, Day 1, 2.5 h post dose | 7.15 [-31.3 to 38.0] | 8.65 [-25.3 to 58.0] | 7.20 [-22.3 to 36.3] | 5.45 [-27.7 to 100.0] | 4.81 [-75.7 to 61.3] | 6.77 [-38.3 to 48.3]
  QTcF, Day before Week 6, 5 min post dose: number analyzed (Participants) | 82 | 78 | 75 | 78 | 83 | 84
  QTcF, Day before Week 6, 5 min post dose | 1.61 [-44.3 to 35.7] | 1.14 [-70.7 to 76.3] | -0.60 [-30.3 to 30.0] | 1.67 [-26.3 to 57.2] | -3.56 [-40.0 to 26.7] | 1.41 [-26.7 to 58.0]
  QTcF, Day before Week 6, 55 min post dose: number analyzed (Participants) | 95 | 91 | 87 | 91 | 92 | 93
  QTcF, Day before Week 6, 55 min post dose | 2.38 [-28.7 to 45.0] | 0.09 [-45.0 to 30.0] | 1.41 [-65.0 to 40.7] | 4.15 [-32.7 to 47.3] | 1.02 [-22.7 to 32.7] | 3.19 [-30.3 to 63.5]
  QTcF, Day before Week 6, 2.5 h post dose: number analyzed (Participants) | 97 | 99 | 90 | 98 | 92 | 100
  QTcF, Day before Week 6, 2.5 h post dose | 4.13 [-32.7 to 40.7] | 0.85 [-64.0 to 51.7] | -0.97 [-55.3 to 48.3] | 1.73 [-44.0 to 49.3] | 0.14 [-31.0 to 33.7] | 2.50 [-29.3 to 44.0]

22. Secondary Outcome: 24-hour Holter ECG - Prolonged QTcF - Male Subjects
Description: 24-hour Holter ECG - Prolonged QTcF - Male subjects.
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5 min, +55 min, and at +2.5 h.
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 63 | 55 | 54 | 58 | 69 | 66
Participants
  QTcF, Day -1, 5 min: Actual value > 450 msec | 1 | 0 | 0 | 1 | 2 | 1
  QTcF, Day -1, 5 min: Actual value > 480 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 5 min: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 5 min: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 62 | 55 | 54 | 57 | 67 | 65
  QTcF, Day -1, 55 min: Actual value > 450 msec | 1 | 1 | 1 | 3 | 1 | 3
  QTcF, Day -1, 55 min: Actual value > 480 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 55 min: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 55 min: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 62 | 54 | 53 | 55 | 68 | 63
  QTcF, Day -1, 2.5 h: Actual value > 450 msec | 1 | 1 | 0 | 2 | 2 | 0
  QTcF, Day -1, 2.5 h: Actual value > 480 msec | 0 | 0 | 0 | 0 | 1 | 0
  QTcF, Day -1, 2.5 h: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 2.5 h: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 62 | 54 | 54 | 56 | 66 | 66
  QTcF, Any post dose time point: Actual value > 450 msec | 3 | 4 | 6 | 4 | 2 | 5
  QTcF, Any post dose time point: Actual value > 480 msec | 1 | 0 | 1 | 0 | 0 | 3
  QTcF, Any post dose time point: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Any post dose time point: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 59 | 51 | 47 | 54 | 67 | 58
  QTcF, Day 1, 5 min post dose: Actual value > 450 msec | 2 | 2 | 3 | 3 | 1 | 4
  QTcF, Day 1, 5 min post dose: Actual value > 480 msec | 1 | 0 | 0 | 0 | 0 | 1
  QTcF, Day 1, 5 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 5 min post dose: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 60 | 53 | 51 | 55 | 68 | 61
  QTcF, Day 1, 55 min post dose: Actual value > 450 msec | 2 | 2 | 3 | 3 | 1 | 4
  QTcF, Day 1, 55 min post dose: Actual value > 480 msec | 1 | 0 | 1 | 0 | 0 | 1
  QTcF, Day 1, 55 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 55 min post dose: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 60 | 53 | 50 | 55 | 68 | 61
  QTcF, Day 1, 2.5 h post dose: Actual value > 450 msec | 3 | 3 | 3 | 2 | 1 | 4
  QTcF, Day 1, 2.5 h post dose: Actual value > 480 msec | 1 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 2.5 h post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 2.5 h post dose: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 59 | 52 | 51 | 56 | 68 | 62
  QTcF, Day before Week 6, 5 min post dose: Actual value > 450 msec | 3 | 1 | 0 | 3 | 0 | 2
  QTcF, Day before Week 6, 5 min post dose: Actual value > 480 msec | 0 | 0 | 0 | 0 | 0 | 1
  QTcF, Day before Week 6, 5 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 5 min post dose: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 60 | 54 | 54 | 55 | 69 | 63
  QTcF, Day before Week 6, 55 min post dose: Actual value > 450 msec | 2 | 2 | 2 | 2 | 0 | 3
  QTcF, Day before Week 6, 55 min post dose: Actual value > 480 msec | 0 | 0 | 0 | 0 | 0 | 1
  QTcF, Day before Week 6, 55 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 55 min post dose: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 61 | 53 | 52 | 56 | 69 | 62
  QTcF, Day before Week 6, 2.5 h post dose: Actual value > 450 msec | 1 | 1 | 0 | 1 | 0 | 3
  QTcF, Day before Week 6, 2.5 h post dose: Actual value > 480 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 2.5 h post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 2.5 h post dose: No prolongation (> 450 msec or > 480 msec or > 500 msec) | 62 | 54 | 54 | 57 | 69 | 63

23. Secondary Outcome: 24-hour Holter ECG - Prolonged QTcF - Female Subjects
Description: 24-hour Holter ECG - Prolonged QTcF - Female subjects.
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5 min, +55 min, and at +2.5 h.
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 58 | 68 | 67 | 65 | 52 | 57
Participants
  QTcF, Day -1, 5 min: Actual value > 470 msec | 0 | 1 | 0 | 0 | 0 | 0
  QTcF, Day -1, 5 min: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 5 min: No prolongation (> 470 msec or > 500 msec) | 58 | 67 | 67 | 65 | 52 | 57
  QTcF, Day -1, 55 min: Actual value > 470 msec | 1 | 2 | 0 | 1 | 0 | 0
  QTcF, Day -1, 55 min: Actual value > 500 msec | 0 | 2 | 0 | 0 | 0 | 0
  QTcF, Day -1, 55 min: No prolongation (> 470 msec or > 500 msec) | 57 | 64 | 67 | 64 | 52 | 57
  QTcF, Day -1, 2.5 h: Actual value > 470 msec | 1 | 2 | 0 | 0 | 0 | 0
  QTcF, Day -1, 2.5 h: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day -1, 2.5 h: No prolongation (> 470 msec or > 500 msec) | 57 | 66 | 67 | 65 | 52 | 57
  QTcF, Any post dose time point: Actual value > 470 msec | 3 | 3 | 0 | 1 | 0 | 1
  QTcF, Any post dose time point: Actual value > 500 msec | 0 | 1 | 0 | 0 | 0 | 0
  QTcF, Any post dose time point: No prolongation (> 470 msec or > 500 msec) | 55 | 64 | 67 | 64 | 52 | 56
  QTcF, Day 1, 5 min post dose: Actual value > 470 msec | 1 | 2 | 0 | 0 | 0 | 0
  QTcF, Day 1, 5 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 5 min post dose: No prolongation (> 470 msec or > 500 msec) | 57 | 66 | 67 | 65 | 52 | 57
  QTcF, Day 1, 55 min post dose: Actual value > 470 msec | 2 | 3 | 0 | 0 | 0 | 0
  QTcF, Day 1, 55 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 55 min post dose: No prolongation (> 470 msec or > 500 msec) | 56 | 65 | 67 | 65 | 52 | 57
  QTcF, Day 1, 2.5 h post dose: Actual value > 470 msec | 1 | 2 | 0 | 0 | 0 | 1
  QTcF, Day 1, 2.5 h post dose: Actual value > 500 msec | 0 | 1 | 0 | 0 | 0 | 0
  QTcF, Day 1, 2.5 h post dose: No prolongation (> 470 msec or > 500 msec) | 57 | 65 | 67 | 65 | 52 | 56
  QTcF, Day before Week 6, 5 min post dose: Actual value > 470 msec | 1 | 2 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 5 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 5 min post dose: No prolongation (> 470 msec or > 500 msec) | 57 | 66 | 67 | 65 | 52 | 57
  QTcF, Day before Week 6, 55 min post dose: Actual value > 470 msec | 0 | 2 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 55 min post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 55 min post dose: No prolongation (> 470 msec or > 500 msec) | 58 | 66 | 67 | 65 | 52 | 57
  QTcF, Day before Week 6, 2.5 h post dose: Actual value > 470 msec | 0 | 1 | 0 | 1 | 0 | 0
  QTcF, Day before Week 6, 2.5 h post dose: Actual value > 500 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 2.5 h post dose: No prolongation (> 470 msec or > 500 msec) | 58 | 67 | 67 | 64 | 52 | 57

24. Secondary Outcome: 24-hour Holter ECG - Prolonged QTcF - Change From Baseline
Description: 24-hour Holter ECG - Prolonged QTcF - Change from baseline.
  Subjects had a 24-h Holter recording before and 24 h after the 1st dose of study drug (Visit 2) and for 24 h before the last dose of study drug (Visit 4). The time-matched values recorded during the 24 h before the 1st dose of study drug on Visit 2 and served as the baseline for the Holter-extracted ECG parameters. The time-averaged baseline score is the average of the Day -1 scores at +5 min, +55 min, and at +2.5 h.
  Results are presented as the number of subjects who had a change from baseline in QTcF of: > 30 msec, > 60 msec, and no prolongation (by > 30 msec or > 60 msec).
Time Frame: Baseline, Day 1, Week 6
Population: Safety population:
  All randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 121 | 123 | 121 | 123 | 121 | 123
Participants
  QTcF, Any post dose time point: Change from baseline: > 30 msec | 19 | 20 | 21 | 20 | 16 | 18
  QTcF, Any post dose time point: Change from baseline: > 60 msec | 0 | 1 | 0 | 2 | 2 | 1
  QTcF, Any post dose time point: No change from baseline (> 30 msec or > 60 msec) | 102 | 102 | 100 | 101 | 103 | 104
  QTcF, Day 1, 5 min post dose: Change from baseline: > 30 msec | 2 | 4 | 9 | 2 | 3 | 4
  QTcF, Day 1, 5 min post dose: Change from baseline: > 60 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day 1, 5 min post dose: No change from baseline (> 30 msec or > 60 msec) | 119 | 119 | 112 | 121 | 118 | 119
  QTcF, Day 1, 55 min post dose: Change from baseline: > 30 msec | 8 | 4 | 5 | 6 | 4 | 5
  QTcF, Day 1, 55 min post dose: Change from baseline: > 60 msec | 0 | 0 | 0 | 1 | 1 | 0
  QTcF, Day 1, 55 min post dose: No change from baseline (> 30 msec or > 60 msec) | 113 | 119 | 116 | 116 | 116 | 118
  QTcF, Day 1, 2.5 h post dose: Change from baseline: > 30 msec | 5 | 12 | 6 | 5 | 6 | 8
  QTcF, Day 1, 2.5 h post dose: Change from baseline: > 60 msec | 0 | 0 | 0 | 1 | 1 | 0
  QTcF, Day 1, 2.5 h post dose: No change from baseline (> 30 msec or > 60 msec) | 116 | 111 | 115 | 117 | 114 | 115
  QTcF, Day before Week 6, 5 min post dose: Change from baseline: > 30 msec | 5 | 3 | 0 | 3 | 0 | 3
  QTcF, Day before Week 6, 5 min post dose: Change from baseline: > 60 msec | 0 | 1 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 5 min post dose: No change from baseline (> 30 msec or > 60 msec) | 116 | 119 | 121 | 120 | 121 | 120
  QTcF, Day before Week 6, 55 min post dose: Change from baseline: > 30 msec | 5 | 0 | 7 | 7 | 3 | 4
  QTcF, Day before Week 6, 55 min post dose: Change from baseline: > 60 msec | 0 | 0 | 0 | 0 | 0 | 1
  QTcF, Day before Week 6, 55 min post dose: No change from baseline (> 30 msec or > 60 msec) | 116 | 123 | 114 | 116 | 118 | 118
  QTcF, Day before Week 6, 2.5 h post dose: Change from baseline: > 30 msec | 6 | 6 | 3 | 6 | 3 | 7
  QTcF, Day before Week 6, 2.5 h post dose: Change from baseline: > 60 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF, Day before Week 6, 2.5 h post dose: No change from baseline (> 30 msec or > 60 msec) | 115 | 117 | 118 | 117 | 118 | 116

ADVERSE EVENTS:
Time Frame: From the first intake of study medication (visit 2, Week 0) until study completion (Visit 4, week 6) or discontinuation.
Description: The safety population was used for the evaluation of treatment-emergent adverse event (TEAEs). The safety population is defined as all randomized patients who received at least one dose of study treatment.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/123 | 0/121 | 0/123 | 0/121 | 0/123
Serious Adverse Events (participants affected / at risk) | 2/121 | 5/123 | 1/121 | 1/123 | 1/121 | 1/123
Other Adverse Events (participants affected / at risk) | 16/121 | 14/123 | 8/121 | 15/123 | 11/121 | 9/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=121) | Treatment B (N=123) | Treatment C (N=121) | Treatment D (N=123) | Treatment E (N=121) | Treatment F (N=123)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=121) | Treatment B (N=123) | Treatment C (N=121) | Treatment D (N=123) | Treatment E (N=121) | Treatment F (N=123)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03084796/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03084796/SAP_001.pdf